# Augmenting Cognitive Training In Older Adults NCT02851511

Document Date: 6/16/2021

#### Protocol - IRB # 201600785

## 1. Project Title

Augmenting Cognitive Training In Older Adults: The ACT Study

## 2. Investigator(s):

## **University of Florida-**

Adam J. Woods, PhD – PI – (Contact PI) Ronald Cohen, Ph.D. - Co-Pl Michael Marsiske, Ph.D. – Co- Pl Mingzhou Ding, Ph.D., - Co-I Christiaan Leeuwenburgh, Ph.D. - Co-I Samuel Wu, Ph.D. - Co-I Eric Porges, PhD - Co-I

#### Staff:

Andrew O'Shea, M.S. Roxanne Razaei, B.A. Jessica Kraft, M.A. Steven DeKosky, M.D. Aprinda Indahlastari, Ph.D. Yunfeng Dai, Ph.D. Yuting Yang Kristin Calfee, B.A.

Alexander Albizu, B.S.

Daniela Carballo, B.S.

Michael Gordon, B.S.

Emanuel Boutzoukas, B.S.

Nicole Evangelista, B.S.

Hanna Hausman, B.A.

Danielle Guess, B.S. Joshua Crow, Ph.D.

Cheshire Hardcastle

Ayden Dunn

Claudia Corbo Kailey Langer

Stacey Alvarez Alvarado

Ruogu Fang

Skylar Stolte

Kyle See

Guanhong Miao

Crysten Repetti

Christina Clarke

Johnna Cesta

Matthew Garrepy

Samantha Pedersen

Nathan Barkdull

#### 3. Abstract:

The current study will investigate methods for enhancing cognitive training effects in healthy older adults by employing a combination of interventions to potentially facilitate neural plasticity and optimize readiness for learning. Adults over the age of 65 represent the fastest growing group in the US population. As such, age-related cognitive decline represents a major concern for public health. Recent research suggests that cognitive training in older adults can improve cognitive performance, with effects lasting up to 10 years. However, these effects are typically limited to the tasks trained, with little transfer to other cognitive abilities or everyday skills. A twophase adaptive randomized clinical trial will examine the individual and combined impact of pairing cognitive training with transcranial direct current stimulation (tDCS). tDCS is a method of non-invasive brain stimulation that directly stimulates brain regions involved in active cognitive function and could enhance neural plasticity when paired with a training task. We will compare changes in cognitive and brain function resulting from CT and ET combined with tDCS using a comprehensive neurocognitive, clinical, and multimodal neuroimaging assessment of brain structure, function, and metabolic state. Functional magnetic resonance imaging (FMRI) will be used to assess brain response during working memory, attention, and memory encoding; the active cognitive abilities trained by CT. Proton magnetic resonance spectroscopy (MRS) will assess cerebral metabolites, including GABA concentrations sensitive to neural plasticity. We hypothesize that: 1) tDCS will enhance neurocognitive function, brain function, and functional outcomes from CT, with combined CT and tDCS providing the most benefit; 2) Effects of tDCS on CT will be maintained up to 12 months following training, and 3) Neuroimaging biomarkers of cerebral metabolism, neural plasticity (GABA concentrations) and functional brain response (FMRI) during resting vs. active cognitive tasks will predict individual response to tDCS. To date, no studies have examined combined intervention strategies using CT or optimization of learning and functional status through facilitation of active versus resting brain states in the elderly. The present study will provide a unique window into critical mechanisms for combating cognitive decline in a rapidly aging US population and possible novel methods for counteracting this looming public health crisis.

#### 4. Background:

**4.1. Public Health / Clinical Significance: 1)** Increased life expectancy has resulted in a marked increase of the older population. **2)** Cognitive changes occur with advanced age that affect functional and health status. **3)** While Alzheimer's and related neurodegenerative diseases cause the most dramatic cognitive disturbances in the elderly, cognitive aging occurs even among people considered to be neurologically healthy. **4)** Even mild neurocognitive disturbances affect people's daily functioning, health status, and quality of life. **5)** Alterations of brain structure and function occur as people reach advanced age, along with cerebral metabolic changes, that are associated with neurocognitive decline. **6)** Our preliminary data suggests that baseline cerebral metabolite (MRS) and functional neuroimaging (FMRI) indices are associated with baseline neurocognitive functioning and predictive of subsequent age-related cognitive decline and brain disturbances. **7)** There is a paucity of preventive and treatment interventions for averting cognitive aging and enhancing cognitive function. **8)** Certain cognitive training (CT) approaches improve specific areas of cognitive performance, although their relative efficacy and mechanisms of action are not well understood. **9)** Most CT approaches do not generalize well to cognitive abilities beyond those being trained or to everyday functional abilities. Efforts are

needed to improve the generalizability of CT. **10)** Methods exist which could feasibly potentiate CT (e.g., tDCS), but they have not been rigorously tested in RCTs.

**4.2. Scientific significance. 1)** While there is evidence that CT can improve cognitive functioning, the underlying mechanisms are not well understood. 2) The efficacy of CT likely is dependent on the plasticity of neural systems. 3) Evidence that certain types of neurochemical, electrical and behavioral stimulation potentiates synaptic plasticity and enhances learning has been demonstrated in laboratory animals. It is important to be able to measure these changes in humans during the course of learning such as that occurring with CT. Yet, in vivo human studies of these effects are difficult for obvious reasons. 4) Functional (FMRI) and cerebral metabolic (MRS) neuroimaging indirectly assess changes in neural plasticity during cognitive tasks. 5) Many open questions exist regarding the brain's structural and functional connectivity in relationship to regional cerebral metabolites. Achieving better understanding of these relationships is important, since cerebral metabolic alterations may contribute neuropathology and perhaps even normal cognitive aging. 6) Extensive research exists for each of these neuroimaging modalities in isolation for various diseases, but multimodal studies employing these approaches simultaneously are less common, particularly in studies of normal aging or CT. 7) Various CT approaches exist, but only a few have been tested and shown to be effective in larger scale clinical trials (e.g., UFOV, dual N-back training). RCTs are needed to test the relative efficacy of these CT approaches, and whether there is value in using them in combination. 8) Brain stimulation may potentiate neural plasticity based on animal studies. Most of these approaches have yet to be tested in conjunction with CT in humans. 9) It is unclear whether optimal CT benefit is achieved by bolstering activation of brain regions necessary for the tasks to be performed. 10) Individual differences exist in the ability of people to benefit from CT. 11) State-of-the-art neuroimaging analysis methods may yield insights into interactions among brain networks/systems, and ways to optimally integrate structural and functional connectivity with cerebral MRS and cognitive outcomes. 12) We will employ state-of-the-art statistical methods, extending predictive modeling and causal inference approaches for neuroimaging.

#### 4.3. Clinical and scientific background.

- **4.3.1.** Cognitive aging and dysfunction affects health status, Quality of Life (QOL), and functional capacity. Brain dysfunction resulting from neurodegenerative disease or other medical condition adversely affects overall health status.<sup>7-11</sup> Even mild cognitive deficits affect QOL, diet, physical activity and other health behaviors, <sup>10,12,13</sup> and are often stronger predictors of health outcomes than other physical factors, <sup>7</sup> but typically receive less clinical attention. Accordingly, cognitive aging has considerable functional relevance.
- **4.3.2. Cognitive training.** Various CT approaches enhance cognitive functioning in the elderly and remediate cognitive disorders. While improvements in cognitive performance are reported in many studies, this research suffers from a lack of well-conducted RCTs designed to determine the specific factors contributing to cognitive improvements. However, several approaches are effective in improving cognitive performance in the context of large RCTs. The ACTIVE study showed that CT improved cognitive performance and resulted in some generalization to other functional abilities.
- **4.3.3. Benefits of cognitive training.** Various CT approaches exist with differing degrees of demonstrated efficacy. While improved cognitive performance is often reported, this research has suffered from a lack of well-controlled RCTs, experimental designs that did not enable the basis for effects to be determined, and limited transfer of training. <sup>14-18</sup> Yet, findings over the past decade (e.g., ACTIVE) suggest that certain CT approaches are effective for enhancing cognitive aging. <sup>17,19-36</sup> Significant cognitive and functional improvements occur in laboratory and homebased CT studies. <sup>19,23,31,37-41</sup> Effect sizes generally exceed d=1.0 immediately after CT, and

even after 10 years ( $\eta^2 > 0.6$ ). In ACTIVE,  $^{22,24,32,36,42}$  people receiving CT outperformed those who were untrained, with normal cognitive aging attenuated. We considered and selected CT approaches based on consensus of our study team (Woods, Marsiske, Edwards, Czaja, et al.), and evidence supporting their effectiveness. Three types of CT training have been particularly effective in studies by our group and others: 1) UFOV; 2) N-back Working Memory; 3) Attentionarousal training, all available in the PositScience BrainHQ suite. Specifically, we will be using eight training programs from the PositScience BrainHQ suite described below.

## Attention/Speed of Processing

- 1. *Hawk Eye* works on visual precision, which helps the brain perceive what is seen quickly and accurately so that it can be recalled better.
- 2. *Divided Attention* requires the brain to focus in on and react to particular details—matching colors, shapes, and/or fill patterns—while at the same time dismissing competing information.
- 3. *Target Tracker* is designed to help build divided attention by requiring participants to track several items moving around their screen at the same time
- 4. Double Decision requires visual search and selective attention to peripheral objects among distractors. Difficulty gradually increases relative to object similarity, presentation rate, and distractor complexity and eccentricity.

## **Working Memory**

- To Do List Training- the brain hears a set of instructions, then uses its memory of those instructions to follow them in order. The instructions get longer and more complex over time at the task, making greater demands on the working memory systems.
- Memory Grid Auditory processing is one of the most important building blocks
  of memory. Only when participants take in information with crystal clarity can the
  brain store it accurately and recall it clearly later. In Memory Grid, the task is to
  match cards representing syllables together.
- 3. Auditory Aces- Participant will be presented with auditory information about playing cards. The information is presented one card at a time. The task is to decide if the current card information matches the card information presented a specific number of steps back in the sequence.
- 4. *Card Shark* N-back working memory task that varies on whether the current target matches stimuli presented 0-n steps before and presentation speed, leading to increased difficulty, 44,45 and age-sensitivity 46.
- **4.3.4. Generalization and functional outcome.** Many CT interventions fail to generate transfer to functional outcomes. Training transfer has been most studied and shown on UFOV. In ACTIVE, ten-year maintenance of UFOV training effects occurred with evidence of substantial transfer at 5 and 10 years. UFOV training resulted in fewer self-reported limitations of everyday activities, higher locus of control 30 and perceived health-related quality of life, he better subjective health, and less depression. At ten years, UFOV-trained people still reported less limitation in daily activities. Self-reported driving cessation and archival accident records indicated lower odds of crashes and driving cessation for UFOV-trained elders at three, five, and ten-years post training. In other RCTs involving greater sustained adaptive CT dosages

(similar to the currently proposed study) superior performance and reaction times were found on a driving-simulator and also for instrumental activities of daily living (look up phone numbers, read pill bottles, etc.).<sup>23</sup> For the other two intervention components, near transfer to other cognitive tasks has been shown. N-back training transfers to matrix reasoning<sup>44</sup> and to sustained attention and self-reported cognitive function in older adults for at least three months post training.<sup>48</sup> Tonic/phasic attention training transfers to spatial selective attention and the temporal distribution of attention (attentional blink).<sup>66</sup>

**4.3.5. Brain stimulation to potentiate training.** Since the pioneering work of Penfield, it has been recognized that sensory, motor and cognitive functions could be altered via electrical stimulation of specific brain regions. In laboratory animals, brain stimulation represented an alternative approach to experimental lesions, enabling both the potentiation and inhibition of neural activity depending on where in the brain stimulation was applied. Until recently, most human brain stimulation studies involved neurosurgically implanted electrodes, which has obvious limitations for general clinical use.

Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation method that alters the sub threshold membrane potential of neurons, facilitates neural plasticity and learning, and increases regional blood flow while modulating local GABA concentrations during stimulation.<sup>69-89</sup> During tDCS, a weak electrical current is applied to the scalp that penetrates skin, bone, CSF and the meninges to stimulate underlying cortical and subcortical tissue. 90-95 tDCS applied to dysfunctional cortical regions improves performance on a variety of cognitive tasks. 96-99 Bilateral tDCS to the frontal cortices improves decision-making, attention and working memory performance in older adults. 100-103 Improvements from a single session of tDCS have been shown to last for up to five years in healthy adults. 104-108 Small pilot RCTs (n=20/group) pairing CT with bilateral frontal tDCS show significant and lasting improvement in older adults experiencing declining cognitive function. 108-112 Maintenance of these tDCS and CT effects have been shown to last beyond one year. 104,105,107,108,110 These studies demonstrate that CT combined with tDCS leads to lasting improvement in CT effectiveness for older adults and patients. Research suggests that increased regional blood flow and decreased GABA concentrations during tDCS facilitate the brain's neural plastic response to paired training tasks. 75,80,83,84,89,113-117 Pairing CT with tDCS to combat age-related cognitive decline may potentially hold great promise for older adults.

- **4.3.6. Age-associated brain changes.** It is well known that with advanced age, humans are vulnerable to neurodegenerative diseases that cause brain pathology, usually evident on post-mortem autopsy. Though less pervasive, neuropathology is also relatively common in elderly adults without documented brain disease. <sup>128</sup>
- **4.3.6.1. Age-associated brain change on structural neuroimaging.** Changes in structural brain volume and morphometry on MRI, along with specific abnormalities, occur with advanced age, particularly when there is vascular co-morbidity. Raz et al. showed cortical and subcortical volume loss of .5 -4% per year across different cortical and subcortical regions in older adults without overt brain disease. Per year across different cortical and subcortical and white matter volume loss across the lifespan in past large international studies. Had, 146, 147, 162-167
- **4.3.6.3. Functional neuroimaging** provides a potentially powerful method for assessing healthy and abnormal brain functioning (see Cohen and Sweet, for a review<sup>168</sup>). FMRI is noninvasive, can be used in conjunction with structural MRI and MRS, and is sensitive to functional brain abnormalities.<sup>153,157,169-179</sup> It holds promise as a biomarker of cognitive aging, neural plasticity, and cognitive improvements following CT. Age-associated alterations in brain activation on FMRI during both rest state and active cognitive tasks have been demonstrated in many past studies. Unfortunately, the clinical potential of FMRI has yet to be fully realized, in part because many different paradigms have been employed across studies. Furthermore, longitudinal change in BOLD response as a function of aging has been examined in relatively

few studies, and almost no large RCTs. Reduced cognitive reserve with aging has been linked to a number of FMRI effects, including HAROLD and PASA. Rolation Change et al. showed that cognitive reserve influences FMRI activation, with a reduced "dynamic range" of BOLD response during tasks relative to rest explaining this effect. Red-190 The concept of dynamic range is both important and useful, and will be discussed in greater detail when reviewing preliminary data (C4).

4.3.6.4. Cerebral metabolites (MRS): Proton MRS, which is sensitive to chemical compounds containing hydrogen, useful for measuring brain metabolites, including N-Acetyl Aspartate (NAA), choline (Cho), myo-inositol (MI), creatine (Cr), and glutamate-glutamine complex (Glx). Our group and others have shown that MRS abnormalities occur among people with a variety of age-related brain disorders, including neurodegenerative disease, cerebrovascular disease, and HIV<sup>191-206</sup>, with reduced NAA and elevated MI associated with cognitive dysfunction and conversion to dementia. Elevated Cho and MI reflect inflammatory processes and glial and cell membrane disturbances, and are differentially associated with cognitive performance, clinical status, and also cortical, subcortical, and white matter volumes on MRI<sup>204-211</sup>. Thus, MRS is predictive of clinically significant neurocognitive dysfunction. 206,208-210 GABA, the brain's principle inhibitory neurotransmitter, <sup>212</sup> is essential for synaptic communication and regulation of neuronal excitability, 213 and neural plasticity. 214-218 It plays a key role in learning and memory<sup>219-235</sup> and modulates other behavioral and affective functions, including executive control and attention. <sup>236-238</sup> Decreased cerebral GABA occurs with advanced age, 219,223,227,230 and GABA dysregulation occurs in neurological and psychiatric conditions. 49,239-<sup>267</sup> GABA delivered to the frontal cortex and hippocampus in animals facilitates cognitive and working memory performance. GABA can now be reliability measured using proton MRS. 5,268-273 based on seminal work by Edden (consultant). 274-278 GABA provides an in vivo biomarker of neural plasticity in brain ROIs important for the cognitive functions to be trained in our study. <sup>276</sup>



Summary and Conceptual Model. Age-associated functional, structural and metabolic brain changes occur, even in the absence of frank neurodegenerative disease. CT holds promise for reducing the adverse effects of cognitive aging, enhancing neural plasticity, cognitive efficiency, functional capacity, and quality of life. In theory, CT benefits could be augmented by coupling it with other interventions that either increase neural plasticity. Yet, relatively few of these approaches

have been tested in RCTs, and the mechanisms underlying their effects are largely unknown. Even less is known about the combined effects of CT with tDCS. Our preliminary data provides strong support for CT to combat cognitive aging, and also for the effects of tDCS on cognition and brain function. We hypothesize that CT leads to improvements in neural plasticity (GABA MRS) and functional brain response (FMRI). In turn, this can lead to improved cerebral metabolic health and structural brain preservation. Coupling CT with tDCS will increase neural plasticity in brain areas important for working memory, focused attention, and executive control, improve effectiveness of CT, and ultimately cognitive health (see Figure 1 for conceptual model).

## 5. Specific Aims:

- **Aim 1.** Determine whether neurocognitive improvement and longer-term functional outcome (as measured by "ecological assessment") are better when CT is coupled with tDCS, an intervention that will increase neuroplasticity and augment training effects.
  - **H1.1.** CT will produce significant improvements on a composite measure of cognitive training performance on the POSIT Science BrainHQ tasks (Posit Composite Score) compared to the treatment control condition. This aim will be assessed at the end of Phase 1.
  - **H1.2.** tDCS combined with CT will produce significant improvements on a composite measure of attention, working memory, processing speed, and executive function (NIH Toolbox Fluid Cognition Composite Score, NIHTB FCCS) compared to the sham treatment control condition. FCCS will serve as the study primary outcome measure.
  - **H1.3.** Near and far transfer of CT and tDCS will occur, as assessed by the UM Functional Battery Composite Index and comprehensive neurocognitive assessment.
- **Aim 2.** Determine whether CT combined with tDCS leads to greater functional and metabolic brain changes (FMRI, MRS). Effects will parallel Aim 1.
  - **H2.1.** Compared to TC, CT will decrease activation in working memory and attentional brain systems (dorsolateral prefrontal cortex, medial frontal cortex, inferior parietal lobe, supplementary motor association cortex), reflecting increased neural efficiency.
  - **H2.2.** Combined CT + tDCS will potentiate these effects.
  - **H2.3.** Cerebral metabolite alterations will occur secondary to CT and tDCS, with long-term increases in GABA and N-acetyl aspartate (NAA) concentrations, and decreased choline (Cho) and myoinositol (MI) concentrations in the frontal cortex and posterior parietal cortex. CT and tDCS will modulate MRS GABA in frontal areas.

**Exploratory Aim.** Examine which baseline factors (e.g., clinical, demographic, neuroimaging, cognitive) best predict individual differences in neurocognitive and functional outcome.

**HE.1.** White matter abnormalities on FLAIR MRI will predict poorer outcome.

undergo neuroimaging at baseline, following CT, and at one-year follow-up.

- **HE.2.** Metabolic-vascular risk factors/disorders (e.g., diabetes) will be predictive of reduced outcome.
  - **HE.3.** Alzheimer's disease risk factors (APOE4 and familial history) will predict poorer outcome.

#### 6. Research Plan:

6.1. Experimental design. This study employs a two-phase randomized clinical trial with 360 participants total across two sites (University of Florida and University of Arizona; 240 at the University of Florida and 120 at the University of Arizona). UF will be the parent site for the study. An initial cohort of 80 participants collected across the two sites will be assigned to one of four conditions as shown in Figure 2. Half of the recruited sample in Phase 1 will undergo CT; the other half will undergo training control (TC). The first interim analysis, to be performed when the first cohort of 80 completes 12-month follow-up (Phase 1), will investigate whether CT is significantly better than TC thereby enabling elimination of the TC condition. CT has previously been established with strong effects on cognitive and functional outcomes. If CT and TC are equally effective, groups will be collapsed at initiation of Phase 2 for planned assessment of adjunctive tDCS effects. If CT is more effective than TC, as previously shown, TC will be eliminated. Data from Phase 1 will also provide important mechanistic insight regarding neural mechanisms of CT vs. a well-matched education training control (TC). In Phase 2, the remaining 280 participants will be randomized to the two CT arms (i.e., eliminating the TC arms). After the remaining 280 participants have completed follow up in the CT arms (including those in Phase 1, total n=360) analyses will investigate the benefit of adjunctive CT+tDCS administration of CT with tDCS. Participants will be assessed at three primary time points: 1) baseline pre-training; 2) post-12 weeks of CT/TC + CT+Sham stimulation/sham; and 3) one year follow-up after all training (see Figure 3 n = 360for timeline). This design will enable longitudinal analyses of CT and tDCS TC+tDCS effects individually and in combination. We will examine CT and tDCS effects TC+Sham on cognitive performance, functional and metabolic neuroimaging measures, and everyday functional abilities. At each assessment, we will obtain clinical and medical history, neurocognitive measures, and neuroimaging (structural MRI, FMRI, MRS). All participants will

- **6.2. Study participants and randomization procedure**. We will recruit 240 older adults (women = 120; age: 65-89 years) at UF. Study participants will consist of healthy individuals who have expressed an interest in taking part in an intervention aimed at optimizing and possibly preserving cognitive functioning and brain health. Web-based permuted block randomization (with block size 8) will be used. In phase 1, each block will have two participants for each arm. In phase 2, each block will have four participants for each remaining arm. We will enroll people with evidence of age-related cognitive decline as defined by performance below the 80<sup>th</sup> percentile on the Cognitive Training assessment. People with pre-existing dementia, neurological brain disease, or who meet criteria for a diagnosis of mild cognitive impairment (MCI) will be excluded.
- **6.2.1. Experimental Design Considerations and Limitations:** CT Approach. The POSITScience BrainHQ treatment program was selected because it 1) provides specific training tasks directed at three essential cognitive domains tied to our aims and hypotheses (attention, working memory, executive control) that correspond with the neurocognitive and functional neuroimaging measures to be studied; 2) is shown to produce significant cognitive and functional improvements with good effect sizes in past RCTs (ACTIVE) with up to 10 year durability and transfer of training to measures of self-reported everyday functioning; 3) provides a "cognitive treatment engine<sup>282</sup>" which alone has a very highly likelihood of yielding significant cognitive and functional improvements, enabling us to test the augmenting effects of tDCS; and 4) is computerized, well standardized, and efficiently implemented.

<u>Combined CT.</u> We selected a combined CT approach rather than testing one specific training task: 1) This would optimize CT treatment effects for this primary intervention, providing a strong and reliable engine of change with which to examine effects of tDCS; 2) This approach enables us to affect several related cognitive functions that are strongly dependent on neural plasticity of the frontal cortex; and 3) This approach would maximize participants interest and motivation versus a single task that could become boring.

**tDCS.** Brain stimulation provides a means of directly augmenting CT effects. tDCS was selected from possible alternatives (e.g., transcranial magnetic stimulation) based on research and data by Woods (PI), including its safety profile, ability to facilitate neural plasticity, and potential for application outside of research settings. Frontal stimulation was chosen based on prior and preliminary studies demonstrating significant impact on attention, working-memory, and other cognitive abilities to be trained during CT. 2mA tDCS was chosen based on prior research demonstrating that this parameter excites, rather than inhibits, activity

in stimulated neurons. <sup>283</sup>

NIH Toolbox. A battery of neurocognitive tests was selected that could be completed in 1.5 hrs for all participants. A battery was selected that would enable optimal assessment of attention, executive functions, and working memory, but would also include some measures of learning and memory, and to a lesser extent other cognitive functions. We use the NIH Toolbox-Cognitive as a core element of this assessment, as it: 1) Can be completed in 30 minutes; 2) Is computerized and well standardized with norms from a large national cohort of older adults; 3) Provides both accuracy and response time measures; 4) Emphasizes the cognitive domains of relevance to the study; and 5) Has been the subject of considerable focus and investment by NIA. This study provides an ideal vehicle for implementing this battery. We supplement the Toolbox with measures to provide more coverage of working memory, attention, learning and memory.

<u>Functional outcome.</u> Since important clinical questions remain with Protocol #201600785

Page 9 of 50

TC+Sham

Cognitively Norma

Baseline Measures

Post CT+tDCS

40 Weeks

1 Year Follow Up

CT+tDCS

CT+Sham

respect to the extent to which CT generalizes to other cognitive abilities and everyday functioning, a set of functional and ecologically derived outcome measures will be used that were developed and used by Czaja (consultant) and her colleagues. Like the NIH Toolbox, this battery is computerized, well standardized with good norms on accuracy and response time from older adults. It taps into important everyday functions such as using an ATM machine and refilling a prescription. See Appendix 2 for detailed manual.

Neuroimaging measures. We will focus on functional (FMRI) and cerebral metabolic (proton MRS) indices for two reasons: 1) These modalities are most linked to and likely sensitive to CT-associated neural plasticity and brain changes; and 2) Changes in these domains are likely to occur over the course of training compared to structural neuroimaging measures. We include active FMRI tasks related to the cognitive functions to be trained, as well as a passive resting state condition to examine the DMN. With respect to MRS, we use a single voxel method to achieve optimal sensitivity and will measure from a single ROI (frontal) corresponding to task and resting state associated brain areas. Along with Creatine (Cr), we will examine cerebral metabolites sensitive neuronal loss and membrane disturbances (NAA, GLx), and proinflammatory processes (Ch, MI). We will also measure cerebral GABA concentrations using a state of art MRS approach that will reflect neural plasticity in ROIs. The MRS indices will be examined for Aims 2.

**6.3. Procedural sequence.** The sequence and flow of the assessments to be conducted at baseline and each subsequent assessment is shown in Subject Timeline.

| Single Subject Timeline | | | | | | | N | /lont | h | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 |
| Phone Screening | | | | | | | | | | | | | | | |
| Consent Form | | | | | | | | | | | | | | | |
| Screening | | | | | | | | | | | | | | | |
| Baseline Measurements | | | | | | | | | | | | | | | |
| Cognitive Training/tDCS | | | | | | | | | | | | | | | |
| Post-CT Measurements | | | | | | | | | | | | | | | |
| 1 Year Follow-Up Measurements | | | | | | | | | | | | | | | |

| Study Timeline | Yea | Year 1 | | | Year 2 | | | Year 3 | | | Year 4 | | | | Year 5 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | 3 | 6 | 9 | 12 | 3 | 6 | 9 | 12 | 3 | 6 | 9 | 12 | 3 | 6 | 9 | 12 | 3 | 6 | 9 | 12 |
| Project Start-Up | | | | | | | | | | | | | | | | | | | | |
| Recruitment/Screening | | | | C1* | | | | | | | | | | | | | | | | |
| Baseline Measurements | | | | C1 | | | | | | :C2: | | | | | | | | | | |
| Cognitive Training/tDCS | | | | | C1 | | | | | | C2 | | | | | | | | | |
| Post-CT Measurements | | | | | | C1 | | | | | | C2 | | | | | | | | |
| 1 Year Follow-Up Measurements | | | | | | | | | C1 | | | | | | | C2 | | | | |
| Interim Analysis (IA) | | | | | | | | IA | | | | | | | | | | | | |
| Final Data Analysis | | | | | | | | | | | | | | | | | | | | |

<sup>\*</sup> Notes: 1) Number of participants in Cohort 1 and 2 are 80 and 280, respectively. The allocation ratio for the last cohort depends on results from IA. Measurements = MRI/Neurocog/Functional Outcomes

**Screening Visit** 

| Task | Estimated Time |
|-------------------------------|----------------|
| Informed Consent | 45 |
| Full medical History/rx drugs | 15 |
| MRI screening form | 5 |
| NACC UDS | 45 |

| WTAR | 5 |
|-------------------------------|----|
| BDI | 5 |
| Computer use questionnaire | 5 |
| Vision/color vision/hearing | 10 |
| AD-8 | 3 |
| Cognitive Training assessment | 20 |

## **Assessment Visits**

| Task | Estimated Time |
|--------------------------------------|----------------|
| MRI scan | 60 |
| MRI scan practice | 20 |
| MRI safety questionnaire | 5 |
| NIH toolbox | 45 |
| Computerized functional task | 40 |
| HVLT | 20 |
| Stroop | 10 |
| PASAT | 10 |
| COWA & Animals | 5 |
| Digit Span | 10 |
| Symbol Digit Coding | 5 |
| Letter-Number Sequencing | 5 |
| Trails A&B | 5 |
| BVMT-R | 20 |
| BDI | 5 |
| STAI | 5 |
| PSQI (sleep) | 5 |
| SF-36 | 5 |
| Apathy scale | 2 |
| PROMIS | 2 |
| AUDIT-10 | 8 |
| DAST-10 | 5 |
| UCLA loneliness | 3 |
| Social Network Scale | 5 |
| CALCAP | 8 |
| IADL Questionnaire | 5 |
| Expectancy Questionnaire | 5 |
| Driving Questionnaire | 10 |
| 10 meter walk test | 5 |
| Abbreviated Medical History/rx drugs | 10 |
| Cognitive Training Assessment | 20 |

We will inform potential participants about the study, and facilitate the informed consent process using the IRB approved ICF. We will then screen for inclusion/exclusion criteria and schedule them for baseline evaluation. All assessments are identical otherwise. Assessment visits will be split over a two-day period, to reduce participant burden and ensure quality data collection.

**6.4 Cognitive Training.** CT will involve sixty sessions over 12-weeks (40 hours total); this includes ten daily sessions combined with stimulation for two weeks, then one weekly session combined with stimulation for the remaining ten weeks. The remaining 40 sessions will be performed by participants at their home on days they do not receive stimulation. *Training platform.* CT employs an eight component, PositScience BrainHQ suite via its researcher portal (described in section 4.3.3). These tasks are web-based and multi-platform (i.e., Windows, Mac). Participants will be required to have minimum screen sizes and specific viewing distances. The interface masks performance feedback to reduce frustration in the control condition. Study interventionists will provide weekly performance summaries. The rationale and task demands for each component were described earlier (A.3.3). These CT are commercially available (www.positscience.com), with well-documented protocols/manuals (See Appendix 1) and thus not described in detail here. Participants will have computers supplied, with training and orientation sessions and 24/7 support.

**Training control**. The TC condition will serve as a control for the CT condition. TC will involve sixty sessions over 12-weeks (40 hours total); this includes ten daily sessions combined with stimulation for two weeks, then one weekly session combined with stimulation for the remaining ten weeks. The remaining 40 sessions will be performed by participants at their home on days they do not receive stimulation. The duration and frequency of TC will match that of CT. TC involves watching educational videos produced by the National Geographic Channel, which cover a range of topics such as history, nature, and wildlife. Participants will be asked to complete questions on the content of the videos to ensure sustained attention.

**Cognitive Training assessment.** An assessment of performance on the 8 cognitive training tasks will be given at the screening and assessment visits. The assessment consists of ten levels (comprised of the games described in section 4.3.3.) designed to challenge working memory, attention, executive function, and speed of processing. The assessment takes approximately twenty minutes to complete.

6.5. Transcranial Direct Current Stimulation: Bilateral Frontal tDCS: A Soterix Clinical Trials Direct Current Stimulator will apply 20 minutes of 2.0mA direct current through two biocarbon rubber electrodes encased in saline soaked 5cm<sup>2</sup> sponges (8cc of 0.9% saline solution) placed over the frontal cortices at F3 and F4 (10-20 system). Based on our well-established computational modeling workflow (C.4.1), F3/F4 stimulation delivers a broad pattern of frontal stimulation (see C.4.1d). Current inflow will occur on the right (F4), and outflow on the left (F3). Impedance quality will be ≤10kΩ to insure proper stimulation of brain tissue. Sham tDCS: Sham stimulation is performed with the same device and all procedures will be identical except for the duration of stimulation. Participants will receive 30 seconds of 2 mA of direct current stimulation at the beginning of the session. Participants habituate to the sensation of tDCS within 30-60 seconds of stimulation. This procedure provides the same sensation of tDCS without the full duration of stimulation, making it a highly effective sham procedure. Blinding: The device has built in RCT double blinding protocols. Soterix will communicate only with Dr. Wu (Co-I/statistician) to de-identify data for analyses. Physiological Recording: During stimulation sessions participants will be asked to wear a special wristband that will be used to record physiological information such as pulse. Quality Control: We will take a brief set of pictures of the participant's head after the electrodes are placed to make sure that the electrodes are in the correct location. These photos will be used to create a 3D model of the participant's head that will give us accurate information about where the electrodes were placed.

**6.6. Neuroimaging Methods.** We will conduct neuroimaging on a Siemens 3.0 Tesla research dedicated scanner with an existing research agreement. Scanning will take 1 hour to acquire: 1) Structural MRI (T1, FLAIR), 2) FMRI (EPI-BOLD), 3) Proton MR Spectroscopy (MRS). **6.6.1. FMRI paradigms.** We will present the two FMRI tasks (2-Back, UFOV) using E-Prime 2 software (Psychology Software Tools, Inc., Pittsburgh, PA), with the video signal on a screen behind the participant's head. The screen is viewed through a double-mirror attached to the head coil. An MR-compatible piano-key response box attached to the stimulus presentation

**2-Back.** This task will measure brain changes due to our N-back training. We will assess verbal

computer will collect performance data. We will apply a cushioned-pillow head stabilizer to



minimize head movement during scanning.

working memory on a 2-Back task, as in past studies<sup>153,157</sup>. Consonants are visually presented briefly with a small rest period between each. Participants determine if each stimulus is the same or different from previously stimuli, responding by binary button press (yes vs. no). Executive control, phonemic

buffering, and sub-vocal phonemic rehearsal are required. 0-back and 2-Back conditions are alternated in a block design with two 5-minute runs of eight blocks (consonant lists), with four blocks of the 0-Back and four blocks of the 2-Back. *0-Back:* Four blocks of nine consonants of random case and order (33% targets). Yes-no responses are made if targets that match stimuli occurring two earlier. 2-Back: Four blocks of 15 consonants (33% targets) will be pseudorandomly presented across the visual field. Accuracy and RT are recorded.

<u>Useful Field of View.</u> This task will measure brain changes due to alterations in attention and decision-making processes due to BrainHQ Double Decision and Freeze Frame training. We will assess attentional and decision-making processes on a scanner adapted event related UFOV task that requires participants to simultaneously apprehend the identification of a centrally located target (car or truck) and the location of a target (car) among a parametrically manipulated array of distractors (0-47 distractors). Following a visual mask, participants then make a two-alternative forced choice (correct or incorrect) decision based on whether both the central target and distal target (without distractors) are identical to what was seen in the prior display (Figure 17). Two five-minute blocks of 56 trials are presented. Accuracy and reaction times are recorded. Jitter prior to stimulus presentation and response probe allows contrasts assessing unique activation associated with attentional and decision-making brain regions, providing mechanistic insight into cognitive training effects.



**Resting State.** Participants will also be asked to rest for 6 minutes while functional data is being collected to assess resting state activation.

**6.6.2. Proton Magnetic Resonance Spectroscopy (MRS):** GABA-edited spectra will be acquired using the MEGA-PRESS experiment, from a 3x3x3 cm3 voxels (medial frontal). Spectra will be analyzed using Gannet and LCModel to assess cerebral metabolites and neurotransmitter concentrations.<sup>295</sup>. <sup>412,413</sup>

- **6.6.3. Structural MRI.** High-resolution whole brain axial gradient-echo MPRAGE 3-D T1weighted images will be acquired for volumetric and cortical thickness analyses and FMRI localization. Analyses: Volumetric indices will be obtained for total gray and white matter, FreeSurfer ROIs<sup>296-298</sup>, and a priori ROIs (MRS, FMRI).
- 6.7. Neurocognitive Assessment: Assessments will include a neurocognitive battery (see Table 7). The battery consists of standardized, well-established neurocognitive measures with strong reliability and validity 304. For cognitive measures with functions assessed see Table 7 below. Our goal is to assess global cognitive ability (NIH-Toolbox: cognitive module), and specifically attention-executive functions, working memory, processing speed, and memory. These are domains affected by aging<sup>24,31,146,305-314</sup> and will also tap the domains assessed by FMRI (Aim 2).

| Table 7. Neurocognitive Assessment | |
|------------------------------------|------------------------|
| HVLT | Verbal Learning/Memory |
| Stroop | Attention/Executive |
| Trail Making A & B | Executive |
| COWA & Animals | Verbal Fluency |
| BVMT | Visual Memory |
| Symbol Digit Coding | Processing Speed |
| Letter Number Sequencing | Working Memory |
| PASAT | Working Memory |
| Digit Span | Working Memory |
| NIH Toolbox Subtests: | |
| * Dimensional Card Sort | Executive |
| * Flanker | Attention/Executive |
| * Picture Sequence | Episodic Memory |
| * Picture Vocabulary | Language |
| * Oral Reading | Language |
| * Pattern Comparison | Processing Speed |
| * List Sorting | Working Memory |

- 6.7.1. Functional Outcomes. A touchscreen computer-based functional assessment tool will be used to measure tasks like medication management, ATM banking, prescription refill via voice menu. Task difficulty can be varied and real-time efficiency and accuracy data are collected; the measure is highly correlated with component cognitive abilities targeted in this study<sup>315,316</sup>. See Appendix 2 for a detailed manual.
- 6.7.2. QOL and PROMIS self-reported health assessment. We will administer the Medical Outcomes Study Short Form-36 (SF-36: v. 2.0, a widely used QOL measure), and the PROMIS self report measures at each assessment. The PROMIS measures assess change in selfreported cognitive and physical function. 321 321. Change in self reported physical and mental health status correlate with QOL and mental and physical health status. 322,323 324 These two measures will serve as important assessments of interventions influence on everyday life.
- 6.8. Alcohol and Drug Use Questionnaires. We will administer the Alcohol Use Disorders Test (AUDIT-10) and Drug Abuse Screening Test (DAST-10). These measures will provide Protocol #201600785

valuable information about how drug and alcohol use may alter the overall efficacy to tDCS, cognitive training and education training.

- **6.9. Driving Record Assessment.** Driving records will be requested following the completion of the intervention; records will be requested at 5 years post intervention and at 10 years post intervention. These records will allow us to examine real world driving outcomes. The driving record assessment is optional (the participant choses to consent to this portion or not at screening). Participants who do not consent to the driving record assessment can still participate in the study.
- **6.10. Walking assessment.** We will administer a 10-meter walk test. This test measures the time it takes participants to walk ten meters in a line. Participants are instructed to walk at their normal pace, as if they were walking down the street. Participants are instructed to use any walking aids they normally use (e.g. cane).
- **6.11. Quality Control.** We will record (with audio and/or video) study procedures for the purpose of ensuring quality data collection. Participants will consent (via a checkbox on the informed consent form) to this recording. Recording will only be done on participants who provide written consent.
- **6.12. Theft Prevention.** This study will be loaning out university computers and other supplies. All university equipment must be returned when the participant completes or withdraws from the study. In the event university equipment is stolen we will be required to file a police report with local authorities. We will make copies of the participant's driver's license when they are provided university equipment. Having a copy of the driver's license provides us with needed information in the event of lost or stolen university property. This procedure is described in the informed consent form. As a driver's license is protected health information it will be kept separate from any de-identified data.
- **6.13. Transportation.** Certain potential participants may lack reliable transportation to the study sites. When possible study staff may transport willing participants to the study sites using a vehicle owned by the Department of Clinical and Health Psychology. All study staff will follow the procedures and regulations for operating University owned vehicles as described by UF Environmental Health and Safety at: <a href="http://www.ehs.ufl.edu/programs/insurance/automobile/">http://www.ehs.ufl.edu/programs/insurance/automobile/</a>

To facilitate transportation to and from the study site Uber Health may be used if the participants desire to have transportation provided. All costs associated with Uber Health will be covered by the study; the participant will not have any cost associated with the Uber Health travel. The option to have travel provided will be offered to all potential study participants within a 40 mile radius of the study site as costs outside of a 40 mile radius will not be feasible with the current travel budget.

Uber Health offers a HIPAA compliant service designed specifically with enhanced ease and privacy in mind for those using the service. Participants will not need to have any account associated with Uber and study staff will coordinate the whole process. The Uber driver will send the participant a text when they are about to arrive at their location, however, the participants personal phone number will not be revealed and instead a covert masking of numbers is provided by Uber to allow the driver and passenger to communicate without revealing their personal phone numbers. If participants do not have or use mobile phones the study coordinator can help coordinate the pickup.

**6.14. Payment.** Participants will receive \$75 in gift cards at the end of each of the three MRI sessions to compensate them for their time and effort.

If participants are traveling from more than 20 miles away (one-way) to the study location they will receive an additional \$10 compensation per study visit. If they attend all study visits they will receive an additional \$270 in compensation for travel. If participants live less than 20 miles away they will receive no additional compensation for travel. If participants are utilizing Uber Health for transportation they will not receive the additional \$10 per visit compensation.

**6.15.** Notification of Participants for Cognitive Findings Leading to Study Exclusion. The Montreal Cognitive Assessment (MoCA) serves as a brief global dementia screening tool commonly implemented in clinical practice. Any participant falling below the 1.5 SD norms (adjusted for age and education) would screen fail in the ACT study, as per current criteria. If this occurs, the participant will first be contacted via phone call by the study physician (Dr. DeKosky) and then provided with a letter from the study team describing their reason for screen fail and encouraging them to follow up with their primary care physician (the letter and phone call template are submitted in miscellaneous attachments in the myIRB system). The procedure for implementation will be built into our RedCap data system such that any person meeting this criterion will trigger an email to the site PI and site physician alerting the team to follow up with the participant and to provide the phone call by the study physician and a letter notifying the participant.

## 6.16. COVID-19 Adjunctive Study

## 6.16.1 Background

In early 2020 the COVID-19 pandemic reached the United States, and has been subsequently spreading rapidly throughout the state of Florida. The pandemic has brought about an exceptional number of public health ramifications. The most striking public response has been to push for a quarantining of exposed, or likely exposed, citizens and a general practice of 'social distancing' for the masses. Additionally, public places frequented by older adults, such as churches and community centers, have been closed leaving an unprecedented number of older adults shuttered in. It has been almost unanimously found that social isolation is a major health problem for older adult populations living in the general community (Nicholson 2012). There currently is a unique opportunity to investigate an enforced social isolation that affects older adults of all demographics. In this study we will record and investigate the outcomes of social isolation for older adults as well as analyze the individual factors that contribute to certain outcomes.

We have a unique set of circumstances where older adults are being forced to remain in their home and away from people indiscriminately. This relative uniformity in social isolation in response to a significant, state-wide crisis allows us to observe the effects of the pandemic on the wellbeing and daily life of older adults, even in adults who might otherwise not experience social isolation in their lifetimes. With such a wide array of people affected we can investigate individual responses to the crisis by looking at a variety of factors as well as track the responses over time.

## 6.16.2 Specific Aims

The following aims will be accomplished using cognitive tests and psychosocial questionnaires in an older population during the immediate COVID-19 pandemic and aftermath:

Aim 1—Assess the current consequences of the COVID-19 social isolation in comparison to pre- COVID 19.

- H.1.1 Social isolation resulting from the COVID-19 pandemic will result in an alteration in cognition, daily living, mental health, and wellbeing in an older adult population.
- Aim 2—Monitor and record changes in the older adult population throughout and following the COVID-19 pandemic and social isolation.
- H.2.1. There will be distinct variations in individual responses to social isolation resulting from the COVID-19 pandemic and there will be observable characteristics that contribute to the differences in response.

#### 16.6.2 Research Plan

**Study timetable and logistics.** Due to the rapidly evolving situation our aim is to administer the study measures as soon as possible pending IRB approval. All adjunctive administrations will be completed with no in person contact via online surveys and telephone calls. At the final COVID-19 assessment time point participants will be asked to complete an in person visit where MRI and blood draw will be done.

Experimental design. Participants will complete the same set of tasks several times starting with acute administration 1, followed by monthly repeats for 6 months, with a final assessment at 9 months following the first. A total of 8 assessments will be completed. Participants will be asked to complete one in person visit at the final COVID-19 time point. At this visit MRI will be conducted to examine possible neurological consequences of social isolation from the ongoing pandemic. Only resting state functional and structural scans will be done as to not impact functional measures of the main study. The MRI will last around 1 hour (see measures section below for additional details regarding the MRI). At this final time point we will also draw a small amount of blood with the aim of conducting COVID-19 antibody testing. COVID-19 antibody testing will allow better classification of previous COVID-19 positive participants. Blood will be collected by a trained phlebotomist in a biosafety level 2 lab at the McKnight Brain Institute and processed in a biosafety level 3 lab. Upon request participants will be provided with their COVID-19 antibody results.

**Participants.** A strength of this proposed adjunctive study is that baseline (pre-COVID-19) data has already been collected on the ACT study sample. This adjunct will allow us to collect additional information in willing participants without interfering with the main study aims. Participation is completely voluntary and in no way affects participation in the main ACT study.

**Recruitment.** Participants who have enrolled in the ACT study will be contacted by phone to assess interest in this adjunctive study. Due to the timing of current events,

we aim to contact all current participants within 30 days of revision approval. However, we will continue to recruit those who we have been unable to make contact with until the PI deems that it is no longer fruitful. Only participants who have been enrolled in the main study prior to March 16, 2020 will be asked to participate in the COVID 19 adjunct. To supplement phone recruitment we will mail letters to eligible participants.

*Inclusion/Exclusion Criteria.* Only participants who have previously provided written informed consent to participate in the ACT study will be contacted. The only additional inclusion criteria is a willingness to participate in the adjunctive measures.

Measures. Adjunctive measures will be conducted via a combination of telephone and REDCap online survey responses. Self-Report questionnaire measures will be completed by the participants using REDCap. An email will be sent to participants with the link to the REDCap survey for them to complete. Cognitive assessments will be completed via telephone and entered by research staff into REDCap. For participants without internet or computer access an option will be provided to complete all measures via telephone. In total each assessment will last around 1 hour. See the table below for an estimate of the time each measure will take. All measures have been previously approved to be completed in the main ACT study with the exception of newly created COVID-19 specific questionnaires. We will be conducting an additional MRI at the 9-month COVID-19 time point.

**MoCA**: A version of the MoCA without visual elements will be completed over the phone. The MoCA is a cognitive screening measure. We will use all three versions of the MoCA in a counterbalanced order over the 8 assessments to limit test-retest effects.

**UDS Number Span:** This measure assesses working memory by asking participants to remember a series of digits and to repeat them in forward and backward order.

**Alcohol Use Disorder Identification Test (AUDIT)**: This measure is a widely used self-report questionnaire designed to assess alcohol use. Alcohol use is common in adult populations and this measure will allow us to quantify use, potential impacts of use, and relate it to stress, individual differences in stress and response to the COVID-19 pandemic.

**Beck Depression Inventory (BDI)**: Symptoms of depression may be a relevant factor in response to uncertainty and social unrest.

**Pittsburgh Sleep Quality Index (PSQI)**: Sleep problems are common. This can impact emotional status and cognition, including sustained attention. Thus, we have selected a measure that assesses sleep quality.

**State-Trait Anxiety inventory (STAI)**: Subjects may experience increased anxiety as a result of the turbulent circumstances surrounding the pandemic.

**UCLA Loneliness Scale**: Designed to measure one's subjective feelings of loneliness as well as feelings of social isolation.

**PROMIS Cognitive Scale**: Assesses a person's perception of cognitive function in areas such as concentration, memory, and mental acuity. Cognitive functions have been known to diminish in periods of extreme stress, which could be aroused as a response to the COVID-19 pandemic.

**PROMIS Physical Function Scale**: Assesses a person's perception of their ability to perform daily activities of living such as chores around the house or carrying groceries.

**Social Network Scale**: Assesses participants' social networks, such as the frequency, time, and number of people they communicate with on a regular basis.

**Medical Outcomes Study Short Form-36**: Self report questionnaire that assesses a variety of functional health outcomes.

Apathy Scale: Measures self-reported feelings of apathy.

**COVID-19 Questionnaire:** Self report questionnaire that assesses the impact of COVID -19 in areas such as a participant's health behaviors, psychological wellbeing, and employment.

**Pet Questionnaire:** Assesses the influence of animal companions during self-isolation.

**Medical Changes Questionnaire:** Assesses any change in medical conditions, such as the worsening or appearance of new health problems.

MRI: We will collect structural T1 images, FLAIR (white matter hyper-intensities), resting state fMRI, diffusion-weighted imaging (white matter integrity) and magnetic resonance spectroscopy (cerebral metabolism). With emerging concerns that COVID attacks the central nervous system, these data will be important for understanding the impact of COVID on brain health in older adults. When compared to each participants most recent ACT MRI, these data will be invaluable for quantifying the impact of COVID-19 on brain health.

#### Estimated time of Online/Phone assessments

| Task | Estimated Time (Minutes) |
|-----------------|--------------------------|
| MoCA | 10 |
| UDS Number Span | 10 |

| AUDIT | 8 |
|--------------------------------|----|
| BDI | 5 |
| PSQI | 5 |
| STAI | 5 |
| UCLA Loneliness Scale | 3 |
| PROMIS Cognitive Scale | 2 |
| PROMIS Physical Function Scale | 2 |
| Social Network Scale | 5 |
| SF-36 | 5 |
| Apathy Scale | 2 |
| COVID-19 Questionnaire | 10 |
| Pet Questionnaire | 5 |
| Medical Changes Questionnaire | 5 |
| Total | 82 |

6.16.3 **Safety Monitoring.** The current pandemic is likely to result in increased mental health problems among the general population. If participants indicate suicidality on the BDI the study psychologist (Dr. Ron Cohen) will immediately contact them for evaluation and referral for treatment.

**6.16.5 Adjunctive Study Payment.** Participants willing to complete the adjunctive study will receive a \$20 payment for their time for each assessment timepoint. This payment is in addition to any other payment they may receive for the main study. An additional \$30 will be paid for the final visit MRI and blood draw.

## 6.17 Safety procedures for resumption of in person research (June 2020)

Additional COVID precautions for assessment/study visits at the MBI. All surfaces in the lab space will be disinfected before and after each participant. Keyboards, mice, ipad screens, etc. will be disinfected before and after each session. 6 foot distancing will be observed in all sessions. PPE will be worn by the participant and the study staff at all times. AMRIS COVID guidelines will be followed for all MRI procedures (MRI compatible PPE, no additional visitors or personnel in the MRI suite, etc.). All study activities occur within the MBI. The MBI has positioned PPE and sanitization stations throughout the ground floor. Participants will be met outside the building by study staff, provided with PPE, if they do not arrive with PPE, and escorted directly to the study location on the ground floor.

Additional COVID precautions for tDCS. For the tDCS intervention, we are required to apply electrodes on the scalp of the participant. As is already our standard, only disposable electrodes are used for each visit to prevent any potential cross participant contact and electrodes are disposed of in biowaste containers after each session. All study staff wear non-latex exam gloves for all study procedures and gloves are disposed of in bio-waste containers after each session. Headstraps to affix electrodes to the scalp will be disinfected

with Clorox after each use. Measurement of electrode locations requires placement of small marks using either a sharpie or wax pencil to determine the precise location for the electrode on the scalp. Thus, the tip of the pen/pencil makes contact with the scalp. Each participant will be assigned a single sharpie/pencil and it will only be used on that participant (labeled with participant ID). Once the participant has completed all intervention sessions, the pen will be disposed of in biowaste. After each session, the pen tip will be wiped with Clorox for disinfection.

**Additional COVID precautions for Cognitive Training.** Participants are provided a laptop for completion of cognitive training. The laptop surfaces will be disinfected before being provided to the participant. For in lab training sessions, the laptop surfaces will be disinfected before and after each session

6.18 Mechanisms, response heterogeneity and dosing from MRI-derived electric field models in tDCS augmented cognitive training

We will leverage existing multimodal neuroimaging and behavioral outcomes data from the ACT trial to 1) elucidate mechanism of action underlying response to tDCS treatment with CT, 2) address heterogeneity of response in tDCS augmented CT by determining how individual variation in the dose of electrical current delivered to the brain interacts with individual brain anatomical and lesion characteristics; and 3) refine the intervention strategy of tDCS paired with CT by evaluating computational methods for estimating precision delivery of targeted dosing characteristics to facilitate tDCS augmented outcomes. We will employ state of the art MRI-derived computational modeling and machine learning (ML) applied to existing data to 1) create precision individualized computational models of electrical current in the brain from tDCS for all 360 participants in ACT (based in T1 weighted images), 2) determine the characteristics of electrical current calculated from electric current models associated with trial outcomes, and 3) evaluate a computational method for calculating possible precision dosing of tDCS parameters for optimizing trial outcomes in older adults.

To date, all prior trials of tDCS have applied a fixed dosing strategy (e.g., 2mA for 20 min with electrodes at F3/F4 [10-20 measurement system]) in attempts to enhance CT – including ACT. However, prior research demonstrates that individual variability in head and brain anatomy (e.g., degree of atrophy, skull thickness, etc.) significantly alters the spread and intensity of direct electrical current delivered to the brain person to person. The impact of individual variation in electrical current delivered to the brain for clinical outcomes has rarely been examined, and methods aimed at increasing stimulation effectiveness and optimizing readiness to learn are only now beginning to be explored. We will use advanced MRI-derived computational modeling of electrical current from existing MRIs to provide a means for accurately estimating individual differences in tDCS current delivery to the brain in the largest existing sample of participants undergoing tDCS (i.e., ACT) with multimodal neuroimaging data. When combined with state-ofthe-art machine learning approaches and behavioral outcome data (only unblinded once ACT has completed all follow-up visits), precision models of tDCS current will be derived to identify critical stimulation dosing characteristics (e.g., current intensity, direction/path of current) in specific brain regions associated with response vs. non-response to tDCS and CT intervention. These data will not only provide much needed information for determining how individual participant characteristics impact tDCS efficacy, but will also serve as a foundation for future precision medicine applications of tDCS and CT to remediate cognitive decline in older adults and potentially prevent or alter the trajectory towards Alzheimer's disease.

- **Aim 1.** Determine inter-individual variability in tDCS current distribution using MRI-derived finite element modeling.
  - **H1.1.** Variability in neuroanatomy (e.g. increased atrophy, sulcus depth, skull thickness, etc.) will significantly decrease current intensity and alter the pathway/direction of electrical current flow induced by tDCS in the brain.
  - **H1.2.** White matter lesions, as measured by white matter hyper-intensities on FLAIR imaging, will significantly decrease current intensity and significantly alter the direction of electrical current flow induced by tDCS.
- **Aim 2.** Determine critical tDCS current properties and specific brain regions associated with responder vs. non-responder to tDCS and CT intervention using machine learning.
  - **H2.1.** Current intensity and direction will significantly predict response vs. non-response to tDCS and CT intervention on the NIH Toolbox Fluid Cognition Composite Score (ACT primary outcome).
  - **H2.2.** Current intensity and direction within bilateral rostral middle frontal, right superior frontal and frontal pole, and left pars orbitalis regions will most strongly predict response vs. non-response to tDCS and CT intervention.
  - **H2.3.** Current intensity and direction will outperform clinical/demographic characteristics alone (e.g., age, sex, comorbidities, mental health, Alzheimer's disease risk, cognition, etc.) in predicting tDCS response.

**Exploratory Aim.** Evaluate computational methods for achieving precision delivery of dosing characteristics in tDCS.

- **HE.1.** Adjusting tDCS current intensity input into computational models will achieve precision delivery of targeted dosing characteristics.
- **HE.2.** Adjusting electrode locations input into computational models will achieve precision delivery of targeted dosing characteristics.

No new data will be collected from participants to achieve these aims. Only existing data collected with consent from participants in the course of the primary ACT study will be used. These data will be analyzed using advanced analytic methods (computational modeling and machine learning) to achieve all three aims specified in section 6.18.

- **Aim 1.** <u>Dependent measures.</u> The primary dependent measure in Aim 1 is current density computed in individual head models from existing MRIs. Current components will be further quantified as current intensity and direction. <u>Rationale.</u> Computed current density will provide an estimate of tDCS current dose within brain regions unique to each person's neuroanatomy. <u>Outcome analyses.</u> **H1.1.** The regression analysis between current density (dependent variable) and anatomical measures (independent variable) e.g., brain volume ratio, sulcus depth, bone thickness will test the hypothesis that unique current density distribution in each person is significantly affected by individual characteristics in neuroanatomy. **H1.2.** Current characteristics generated from models will be compared between inclusion and exclusion of white matter lesions. A false discovery rate (FDR)-corrected voxel-wise within participants analysis will test the hypothesis that inclusion of white matter lesions in computational models significantly alters current characteristic predictions.
- Aim 2. <u>Dependent measures</u>. The primary dependent measure in Aim 2 is balanced accuracy. This measure provides an overall index of the performance to differentiate responders from non-responders. <u>Rationale</u>. By using this measure, we provide a single performance indicator upon which the **heterogeneity of response** in tDCS augmented CT can be revealed. Much of our preliminary data is based on analyses using this measure. <u>Outcome analyses</u>. All analyses will be conducted with the intent to optimize prediction of tDCS outcome. McNemar test at one-tailed 0.05 significance level will be conducted to determine whether current intensity and direction will outperform clinical and demographic characteristics alone in predicting tDCS response.

**Exploratory Aim.** <u>Dependent measures.</u> The primary dependent measure in the Exploratory Aim is log-likelihood distance measure. Adjustments of electric current intensity and electrodes placement in computational models will be used to minimize the log-likelihood distance measure to the Gaussian Mixture Model of the responders' current distribution.

**Timeline.** Construction of the MRI-derived finite element computational models as described in aim 1 is estimated to begin in January 2021. We estimate approximately 24 months will be required to complete this process. By Q3 2022 the ACT study is anticipated to be completed and access to the currently blinded randomization conditions will be available to complete aim 2 and the exploratory aim.

The additional analyses described in section 6.18 will not impact study participation in any way. The analyses will only use data collected under currently approved study procedures.

#### 7. Possible Discomforts and Risks:

#### Potential Risks.

There are minimal risks associated with participation in this study. The potential risks are as follows:

Magnetic resonance imaging (MRI). MRI is a procedure that allows doctors to look inside the body by using a scanner that sends out a strong magnetic field and radio waves. This procedure is used routinely for medical care and is very safe for most people, but participants will be monitored during the entire MRI scan in case any problems occur. The risks of MRI are:

- The MRI scanner contains a very strong magnet. Therefore, participants may not be able to have the MRI if they have any type of metal implanted in their body, for example, any pacing device (such as a heart pacer), any metal in their eyes, or certain types of heart valves or brain aneurysm clips. A MRI technologist will question participants about any contraindications before they enter the scanner.
- There is not much room inside the MRI scanner. Participants may be uncomfortable if they do not like to be in close spaces ("claustrophobia"). During the procedure, participants will be able to talk with the MRI staff through a speaker system, and, in the event of an emergency, participants can tell them to stop the scan.
- The MRI scanner produces a loud hammering noise, which has produced hearing loss in a very small number of participants. Participants will be given earplugs to reduce this risk, and headphones for added protection.
- If an obvious abnormality is discovered during the participant's MRI scan, they will be
  informed about it by the research team, and will be provided with a copy of the MRI scan and
  we will encourage them to see their primary care physician. MRI will only be done for
  research purposes in this study.
- Participants will be monitored very carefully while in the scanner, and repeatedly checked to ensure comfort.

<u>Transcranial direct current stimulation.</u> Transcranial direct current stimulation is considered safe but a small number of people do experience some side effects. The most common side effects are itching and tingling or mild discomfort at the area of stimulation, and headache. Other possible side effects include dizziness and nausea. Whenever an electrical stimulation is applied to the body, it could possibly cause a seizure or abnormal heartbeat, but this has never occurred with the transcranial direct current stimulation parameters used in this study.

<u>Cognitive Training.</u> There is a risk participants will find cognitive training on the computer challenging, fatiguing, and/or boring. Research staff will explain what to do and how to perform the training tasks tests during an initial study visit. Participants will also have access to a 24-hour help line should they have trouble working with the training computer.

<u>Educational training.</u> There is a risk participants may find ET to be challenging, fatiguing, and/or boring. Research staff will be present to address any concerns. Participants are free to skip any content they find objectionable and refrain from answering any questions that they find uncomfortable. All material presented has been judged appropriate for an educational setting.

<u>Neurocognitive and Functional tests</u>. There is a risk that participants will find cognitive and functional tests challenging, because it may be difficult to remember the things that they are asked to remember or participants may have trouble hearing or seeing some of the sounds and pictures presented on the computer screen. Participants may skip any tests they do not wish to complete. Research staff will explain what to do and aid participants during their study visit.

<u>Questionnaires.</u> There is a risk that participants will find questions on the questionnaires uncomfortable to answer. Participants may skip any question they feel uncomfortable answering.

Participants will be asked questions about previous and current alcohol and drug use with two questionnaire measures (AUDIT-10 and DAST-10). These questions are of a particularly sensitive nature. There is a risk that participants may feel uncomfortable about answering such questions. Like any other part of the study, participants are free to decline to answer anything that they are uncomfortable with.

Other possible risks to participants may include fatigue due to the testing. Should this occur, participants can take a rest-break at any time or may discontinue the testing at any time.

When being tested some people may develop anxiety. If these tests make participants anxious we can stop the testing.

Researchers will take appropriate steps to protect any information they collect about participants. However, there is a slight risk that information about participants could be revealed inappropriately or accidentally. Depending on the nature of the information, such a release could upset or embarrass participants, or possibly affect their insurability or employability.

This study may include risks that are unknown at this time.

Participation in more than one research study or project may further increase the risks to participants. If participants are currently participating in another study using transcranial direct current stimulation or transcranial magnetic stimulation, they will not be enrolled in this study until all external studies are completed.

If participants consent to the COVID-19 ancillary blood draw risks associated with phlebotomy apply. These include discomfort at the site of puncture, possible bruising and swelling around the puncture site, rarely an infection, and uncommonly faintness from the procedure.

### Adequacy of Protection against Risks.

<u>Recruitment and Informed Consent.</u> All study participants will provide written informed consent. Persons will be recruited from the CAM-CTRP research registry, advertisements such as

newspaper, magazine, and bus ads. community outreach, or community agencies. Participants will also be recruited at community events with IRB-approved flyers, and participants will have the option to confidentially provide name, phone number, and email if they wish to be contacted by the study team to determine study eligibility. Contact information will also be obtained through the UF Health Consent2Share registry to identify potential participants. If Consent2Share contacts are interested in hearing more about the study, they will be administered the phone screening. If we are unable to reach potential participants we will leave a phone message (see phone message script) to let them know the reason for our call. If they are interested in hearing more about the study they will be directed to call us back and then administered the approved phone screening after confirming initial interest and addressing any questions they may have. The contact information will be securely stored during the event and immediately stored in the Woods Lab after the event per study data safety management plan. People interested in participating in the study will call the CAM-CTRP study recruitment coordinator. Potential participants interested in hearing more about the study will be provided information about the study. Persons will then indicate their agreement to participate by signing the informed consent document.

Our inclusion and exclusion criteria are designed to minimize risks to participants.

#### Inclusion criteria:

- 1. Age 65 to 89 years; this age group was selected because it is at high risk of age-related cognitive decline and have a sufficiently long life expectancy<sup>319</sup> to participate in the study;
- 2. Evidence of age-related cognitive decline in the Cognitive Training assessment defined by performance below the 80<sup>th</sup> percentile.
- 3. Ability to participate in the intervention and attend training sessions; willingness to be randomized to either treatment group.

Rationale: (1) The age range is selected to include a higher proportion of persons with cognitive deficits. (2) Participants will need to show some form of impairment to be included in the study in order to avoid biasing the study with extremely high functioning individuals. (3) Participants must be willing to perform study activities.

Exclusion criteria: 1) Neurological disorders (e.g., dementia, stroke, seizures, traumatic brain injury). 2) Evidence of cognitive impairment (as defined by NACC UDS performance below 1.5 standard deviations on age/sex/education normative data in at least one cognitive domain). 3) Past opportunistic brain infection 4) Major psychiatric illness (schizophrenia, intractable affective disorder, current substance dependence diagnosis or severe major depression and/or suicidality. 5) Unstable (e.g., cancer other than basal cell skin) and chronic (e.g. severe diabetes) medical conditions. 6) MRI contraindications (e.g., claustrophobia, metal implants). 7) Physical impairment precluding motor response or lying still for 1 hr and inability to walk two blocks without stopping. 8) Currently on GABA-ergic or glutamatergic medications, or on sodium channel blockers. 9) Left-handedness.

Rationale: (1) neurological diseases affecting the brain create obvious confounds that would obscure the study's findings or increase risk from non-invasive brain stimulation (i.e., seizures). (2) The NACC UDS will be used to exclude people meeting criteria for severe dementia, as this study is focused on more mild-moderate cognitive impairment; (3) past opportunistic brain infection, and (4) a history of severe psychiatric illness (schizophrenia, chronic intractable unipolar or bipolar depression) also would directly affect neurocognitive test performance and thus would confound study findings. (5) Unstable (e.g., cancer) and certain chronic medical conditions (e.g., severe obesity) may also confound findings and increase study attrition; (6)

Given that this study requires MRI imaging to address all aims, factors that make MRI imaging unsafe or infeasible for particular study candidates will serve as a basis for exclusion; and (7) Physical limitations are a basis for exclusion based on inability to participate in all study procedures. Excluding people who cannot walk or sit for an hour will reduce problems in the scanner that could confound study findings. (8) GABA-ergic, glutamatergic, or sodium channel blocking medications may alter or block the ability of tDCS to facilitate tissue excitability. (9) Left-handedness complicates the interpretation of FMRI findings.

## Protection against Risk.

Protection against Risk of confidentiality. Information pertaining to research subjects will be obtained from (1) interviews with subjects and (2) procedures described in the "research design and methods" section. All data will be considered confidential according to HIPAA guidelines for personal health information. All participants will sign a combined consent to participate in research and HIPAA compliant confidentiality document approved by the IRB overseeing the clinical recruitment setting (i.e. the University of Florida IRB, and the Florida Department of Health IRB).

Precautions will be taken to ensure that all research materials are inaccessible to anyone other than the investigators, and by ensuring that only qualified and trained individuals conduct the study research procedures. Prior to study initiation, procedures for protecting the confidential nature of participant data collected will be reviewed and all questions or concerns will be clarified at this time. These procedures will be reviewed throughout the study. Staff will be trained and certified in handling human subject information to maintain privacy and confidentiality. Procedures for allowing access to investigators to use this information for research will be under the authority of the PI and will follow HIPAA compliant guidelines for the release of PHI.

Contact information for study participants will be kept in separate files and databases from the research data. This information will be used by the research assistants to send reminders about follow-up times and appointments via phone, email, or mail correspondence depending on the participant's preference. Research assistants may contact study participants via phone, email, or mail to provide directions to the study site or answer general questions or concerns about the study. In order to avoid participants who are lost to follow up, we will contact study participants periodically between their 3 month post intervention visit and their one year follow up visit at approximately 3 month intervals. We will send a letter and/or email to participants who we are unable to contact via phone to see if their contact information has changed. The information will only be kept on computers or devices that are both password protected and encrypted. Any written forms will be kept in locked file cabinets or locked briefcases. None of the research data in the central database will have participant identity information. No results will ever be reported in a personally identifiable manner. All research data will be entered directly into a web-based survey that is maintained by the University of Florida CTSI (REDCap), and the data are encrypted as soon as they are sent in a wireless format. The data will be transferred and stored on secure servers at the University of Florida, with no identifying information. Only de-identified data will be entered into the REDCap database across all sites. A data confidentiality agreement will be signed and filed with the UF IRB before any data are collected at any site.

No survey data will be labeled with the participant's name or other identifying information, but will instead be labeled with a study ID number. Documents linking study ID numbers to identifying information (e.g., name, address, etc) will be stored electronically in a password-protected file. All paper-data with identifying information will be stored in locked file drawers, separate from coded data. Documents linking study ID numbers to identifying information will be destroyed at the end of the study. Documents containing data collected on un-consented

individuals (i.e., screening logs used to avoid approaching the same individual for study enrollment twice) will be shredded daily. All electronic data will be secured and encrypted. Identifying information will not be reported.

Protections of risks related to study questionnaires. To minimize any risks related to emotional responses to questionnaires, persons will be informed about the types of questions included in the surveys, which are similar to the types of questions persons might be asked by their doctor in a clinical setting.

Protection of risks related to tDCS. To minimize risk associated with tDCS, participants will be monitored throughout stimulation sessions and asked to report any discomfort. If scalp sensation is uncomfortable, stimulation will be stopped. In the event of a headache, stimulation will be stopped. All tDCS sessions will be administered and continually supervise by a trained experimenter. The above symptoms have only been reported when participants are actively being stimulated. However, to assess for any symptoms occurring during the 24 h interval between stimulation sessions, we will administer a brief symptom screening questionnaire at the beginning (symptoms in the past 24 hours) and end of each session (symptoms during stimulation). tDCS has not been shown to cause seizures nor lower the seizure threshold in animals. There are no reports of seizure induced by tDCS in human participants in the literature. However, this may not be true for epilepsy patients, whose seizure threshold rates are likely abnormal. Prior history of neurological disorders is an exclusionary criterion for our study and thus no participants will have a history of seizure.

Protection against risks associated with neuroimaging. MRI is widely regarded as a safe, noninvasive procedure for visualization of brain tissue in both adults and children. Prior FMRI studies by our group and by other groups document the innocuous nature of these procedures. Prior to study participation, all participants will be informed of the MRI procedure during the informed consent/assent process. The proposed study will be performed on an FDA approved Siemens 3 Tesla scanner located at the Advanced Magnetic Resonance Imaging and Spectroscopy (AMRIS) research facility at UF. There are no known long-term effects of MRI procedures on the body. The FDA Information Sheets, Food and Drug Administration, October 1995, p. 79, lists as a non-significant risk device, "Magnetic Resonance Imaging (MRI) Devices within FDA-specified parameters." This study satisfies those parameters. The 3.0 tesla MR scanners meets FDA parameters for field strength, gradient switching, and RF power deposition for all FDA-approved acquisition schemes including echo-planar imaging. In addition, this research protocol involves the use of an FDA-approved acquisition scheme, or the power deposition of experimental acquisition scheme proposed meets FDA parameters as verified on a phantom using the power monitoring system installed on the MR scanner. Both Dr. Woods and trained MRI staff will check for exclusion criteria. The main MRI-related risks include: (a) sensitivity to the loudness of the MRI machine - all subjects will be given and must wear ear plugs; a squeeze-ball and microphone will be provided so that they may stop the testing if they become uncomfortable or anxious at any time; (b) claustrophobia - subjects will have the opportunity to practice in a simulator and to become as familiar and comfortable as possible before commencing the experiment. In addition, they will be given the opportunity to examine the scanner before the tasks starts. The study will be ended early if the space is a problem for them; no medications (e.g., benzodiazepines or tranquilizers) will be offered to them; (c) lightheadedness when sitting up after lying in the MRI machine - this feeling sometimes occurs but has always gone away in a few minutes. Participants will thus be assisted in getting up to make sure they do not fall; In sum, the MRI neuroimaging procedures pose no radiological or medical risk, given that participants with metal implants susceptible to magnetic heating will be excluded based on standard scanner policies. A small number of people may become anxious

in the small space of the scanner. These individuals will have the opportunity to terminate the scan session. Furthermore, all recruits will be screened for phobias prior to enrollment. There is a medical technologist at the imaging site at all times to insure scanner safety, and neuroradiologists on call as needed. If an abnormality is noted on the structural MRIs by study staff, the PI will provide the participant with a copy of the scan and encourage them to follow up with a neurologist.

Protection against risks associated with neurocognitive tests. The neurocognitive assessments have minimal risk associated with them. Some participants experience stress associated with being tested, though this tends to be quite limited. Breaks will be given in those cases. Research staff that collect data have been trained in the conduct of all cognitive function tests by other senior staff members. Research staff members will be certified in the conduct of the cognitive function tests before they work with study participants.

## **Data and Safety Monitoring Plan:**

The research team will follow the procedures for data safety and monitoring as required by the Institutional Review Board at the University of Florida (UF IRB). The research team will monitor participants for any potential adverse events, and all reported events will be forwarded by the PI to the UF IRB.

A data and safety monitoring plan (DSMP) has been implemented to ensure the safety of all participants involved in the study and to ensure the validity and integrity of the data. The primary goal of the DSMP will be to monitor the progress of the study and safety of participants and if necessary, recommend modifying the study or terminating the study as appropriate.

- The PI's will be responsible for coordinating activities of the DSMP, including:
  - Lab Meetings twice per month, to discuss participant involvement in the study, and any issues that have developed or need revision
  - Safety concerns
  - Data Storage and safety
  - Participant safety
  - Outcome data
  - Data quality
  - Integrity
  - Intervention efficacy
  - Recruitment
  - Performance

Both the PI and the study staff will review and examine reports of adverse incidents immediately, and make reports to the IRB as necessary for any and all of the following situations:

- Serious and non-serious adverse events that may occur
- Suspicion of scientific fraud or misconduct
- o Any other issues which may warrant protocol changes or modifications.

<u>Procedure for collection and storage of data.</u> A number of quality control procedures will be used to ensure the validity and integrity of the data and the safety of all participants involved in the study. Relevant data and safety information obtained on each study participant will be verified against the original source documents by the primary study coordinator and any

identified discrepancies will be reviewed at these meetings. The primary goal of these meetings will be to monitor the progress of the study and safety of participants and if necessary, recommend modifying the study or terminating the study as appropriate.

All identifying information will be archived in Dr. Cohen's and Woods neuroimaging laboratory within the Center for Cognitive Aging and Memory. Imaging data will undergo several levels of processing, and all raw and processed data will be archived on a University password-protected server in password-protected folders and files. Only study staff will have access to these files. The self-report data will be double entered using the RedCap Data System. This system signals the user when an out-of-range value is entered. All data entry is then verified via double-entry, with the program signaling mismatches with the original entry. Next, computer-generated reports of variable frequencies and subject lists will be reviewed, leading to possible corrections to coding or entry. After checking for accuracy of data within a given group, data will be stored in

Location and logistics of data collection. All procedures involving human subjects will be performed at facilities of the UF Health Care System. Neurocognitive testing and training will be performed at the clinical research unit of the Center for Cognitive Aging and Memory with an ancillary location at the Village at Gainesville. Several clinical research examination rooms are equipped and dedicated to neurocognitive and functional assessment, and contain all necessary computers and test materials. Storage of neuroimaging data backup will occur at the CAM Neuroimaging Laboratory. Neuroimaging will take place at the AMRIS facility of the McKnight Brain Institute.

the password-protected folders along with the imaging data.

Sharing of data from collaborating sites. Due to the multi-center design of the study, data will be shared with the University of Florida from a collaborating site, the University of Arizona. The collaborating site will send fully de-identified data. Data transfer will take place using the secured infrastructure of the University of Florida RedCap system for questionnaire data. De-identified raw neuroimaging data will be transferred to UF using the Secure File Transfer Protocol (SFTP) onto UF Dropbox servers. A data confidentiality agreement will be signed and filed with the UF IRB before any data are collected at any site.

Storage of collected data. All electronic data are stored in password protected, secured computer systems. All paper data will be stored in a locked file cabinet. Data will only be removed when coded, entered, or audited. Only the participant's study identification number will appear on any data forms. Only the PI, the Co-Is, and the RAs will have access to the completed data forms and electronically stored data. All data are considered part of the participant's confidential record. Data collected from research participants will be stored in a secured, password protected computer file that is separate from network systems. All paper data (e.g., subject contact information, consent forms, etc.) will be placed in a locked file cabinet within 24 hours of their acquisition as designated by the study's RA. All data will remain confidential. Data entry requirements. The data entry system will require a login identification and password in order to gain access to the data. Where appropriate, validation and range rules will be applied to the actual entry fields. Only the PI and Co-Is will be able to view the data in its raw state.

<u>Audit/verification of entered data.</u> All data designated as primary outcome data will be subject to a 100% cross-referencing between electronic and paper forms. This audit must have an error rate less than 1%. If the verification fails the audit, all data will be re-entered, the original computer files discarded, and the newly re-entered data audited. This process will continue until the audit no longer exceeds the maximum allowable error rate. All audits will be supervised and documented by the PI.

<u>Data management and analysis</u>. Our research team has substantial experience in the design and implementation of data management procedures that provide accurate recording and storage of data, participant confidentiality, and timely analysis. Based on our past experience, we believe that our major data management and analysis needs for the proposed project can be met by using a high-end PC, equipped with the latest version of SPSS for Windows and appropriate spreadsheet programs. All data files are automatically backed-up daily.

<u>Data quality control</u>. All staff involved in data collection will be trained and certified to ensure their competence, and re-certified periodically throughout the study as we have done in similar trials. Data will be collected and numerically coded using pre-tested electronic entry forms. At the time of collection, there will be initial clerical review of all data for accuracy and completeness. Every effort will be made to ensure that missing data are kept to a minimum. Data entry programs with range checking and response validation will be used for all data entered. Under supervision from the PI, the data manager will conduct error checking procedures and preliminary analyses on all data to ensure their accuracy. The RAs will be trained to avoid omissions in data entry and computer entry protocols will be programmed to avoid accidental skipping of question items. We believe that the quality control system to be used will ensure a complete and accurate database, and maximize the likelihood that the intervention will be delivered correctly and efficiently. As we have done in prior studies, a manual of procedures will be developed during the initial study start-up period that explicitly describes the specific procedures related to intervention delivery, data collection, and quality assurance.

<u>Frequency of data review.</u> Relevant data and safety information obtained on each study participant will be verified against the original source documents by the primary study coordinator on a bi-weekly basis. As noted above, any identified discrepancies will be discussed with the Principal Investigator and reviewed at weekly meetings.

Measurement and reporting of participant accrual and adherence to eligibility criteria. Review of the rate of participant accrual, adherence to inclusion/exclusion criteria will occur weekly during the recruitment phase and then every month to assure that participants meet eligibility criteria and ethnic diversity goals outlined in the grant proposal.

<u>Safety Review Plan</u> Study progress and safety will be reviewed twice per month (and more frequently if needed) by the principal investigator. An annual report will be compiled and will include a list and summary of AEs. In addition, the annual report will address (1) whether adverse event rates are consistent with pre-study assumptions; (2) reason for dropouts from the study; (3) whether all participants met entry criteria; (4) whether continuation of the study is justified on the basis that additional data are needed to accomplish the stated aims of the study; and (5) conditions whereby the study might be terminated prematurely. The IRB and other applicable recipients will review progress of this study annually.

<u>Final storage of paper data.</u> All paper data (e.g., consent forms) may be scanned, and will finally be housed at a facility that specializes in the storage of medical/ research information. The destruction date of these files will be at least 7 years from the termination of the study and will be authorized by the Principal Investigator of the research study.

Access to cleaned computer data. Once the study is complete, and all data have been collected, entered and passed the audit process, the data will be available to the Principal Investigator and his designates for analysis. Only the Principal Investigator can give permission for the release of aggregated study data. No confidential information may be released without

the express written consent of the study participants. Only copies of the finalized data will be released. The original data file will remain in its pristine state.

<u>Description of plan for safety monitoring.</u> Protection of participants from risks related to the study is of paramount concern.

Monitoring physical health and safety. All assessment visits will be conducted at a central location and all testing sessions will be conducted and supervised by a trained and certified research staff that will monitor potential adverse experiences and symptoms. At each visit, participants will be asked to report any adverse events they have experienced since their last visit. Immediate medical treatment will be provided for any illness or injury resulting from this study. Trained nursing staff members are present in the research center at all times, and a physician will also be available to evaluate the participant if needed.

In addition to the assessments conducted at in-person study visits, participants will be asked about any adverse events, including itching, pain, nausea, headache, etc. they have had. Participants will also be asked about their mood, including depressive symptomatology, and other health related activities (i.e., physical activity), as well as general health status. Based on reported symptoms, participants may be asked to come in for an additional follow-up assessment visit with one of the healthcare professionals on the study team (i.e., physician or psychologist) for further evaluation of their symptoms. Based on information obtained at this visit, participants will then be referred for follow-up assessment and/or treatment with the appropriate healthcare provider.

Monitoring mental health and safety. Any participant who endorses clinical levels of any psychiatric disorder or who endorses suicidality will be referred to Dr. Cohen, study psychologist, for further follow-up assessment. The psychologist will then provide a recommendation regarding the appropriate course of follow-up and also advise on whether it is safe for the participant to continue in the study. If a participant is found to be actively suicidal with a plan and/or intent, they will be escorted immediately to the emergency room at the Shands Hospital at the University of Florida. If safety is an issue, UF security or local authorities will be called for assistance.

## Data and Safety Monitoring Board (DSMB):

A **Data Safety Monitoring Board (DSMB)** is established, with responsibility to monitor all aspects of the study, including those that require access to any masked data. The DSMB and its chair are named and approved by the NIA. It is planned that the DSMB meets by conference call as determined by the DSMB and the NIA. The DSMB has access to all deidentified study data, documents and progress. The Intervention and Safety Committee, **comprised of safety personnel from each site, the Chair, and a representative of the DMAQC** reports to the DSMB for issues related to participant safety.

The DSMB has the following charges:

- Review the study protocol.
- Review data (including masked data) over the course of the trial.
- Identify problems relating to safety over the course of the study.
- Identify needs for additional data relevant to safety issues and request these data from the study investigators.
- Propose appropriate analyses and periodically review developing data on safety and endpoints.
- Make recommendations regarding recruitment, treatment effects, retention, compliance, safety issues and continuation of the study.

• At any time, the DSMB may recommend discontinuation of any component/treatment group of the study

Finally, the NIA makes the final decision on whether or not to accept the DSMB's recommendation about discontinuation of any component of the study. Any serious adverse event that might be due to the study intervention are reported to the DSMB, the IRBs, and to the NIA Project Office. The exact timeline for reporting serious adverse events is determined by the DSMB, IRBs, and NIA.

#### 8. Possible Benefits:

There are well-documented benefits for older adults who participate in cognitive training, including improvement in working memory, attention, and executive functions. Deficits in these cognitive abilities significantly impact quality of life, financial capacity, medication adherence, and mortality in older adults. Those participants randomly assigned to the CT groups may benefit from these effects. Participants assigned to the Education Training Control group may obtain better knowledge about educational facts from the videos, but are unlikely to have the same benefits as those in the CT group. Those participants randomly assigned to the tDCS+CT treatment group may experience further benefit beyond that of cognitive training alone. Benefits to society will include the contribution of novel data regarding the efficacy of neuromodulation methods for enhancing cognitive training effects in older adults. This may help inform treatment protocols in a growing segment of the US population (i.e., those 65 years and older). Data collected from this study will serve as a foundation for larger clinical studies that examine optimized methods for treating aging-related cognitive decline using cognitive training and tDCS. Some participants may not benefit from the study at all.

#### 9. Conflict of Interest:

#### None

- 1. Sumner P, Edden RA, Bompas A, Evans CJ, Singh KD. More GABA, less distraction: a neurochemical predictor of motor decision speed. *Nat Neurosci.* Jul 2010;13(7):825-827.
- 2. Streeter CC, Jensen JE, Perlmutter RM, et al. Yoga Asana sessions increase brain GABA levels: a pilot study. *J Altern Complement Med.* May 2007;13(4):419-426.
- 3. Edden RA, Muthukumaraswamy SD, Freeman TC, Singh KD. Orientation discrimination performance is predicted by GABA concentration and gamma oscillation frequency in human primary visual cortex. *J Neurosci*. Dec 16 2009;29(50):15721-15726.
- 4. Puts NA, Edden RA, Evans CJ, McGlone F, McGonigle DJ. Regionally specific human GABA concentration correlates with tactile discrimination thresholds. *J Neurosci*. Nov 16 2011;31(46):16556-16560.
- 5. Gao F, Edden RA, Li M, et al. Edited magnetic resonance spectroscopy detects an agerelated decline in brain GABA levels. *Neuroimage*. Sep 2013;78:75-82.
- 6. Streeter CC, Whitfield TH, Owen L, et al. Effects of yoga versus walking on mood, anxiety, and brain GABA levels: a randomized controlled MRS study. *J Altern Complement Med.* Nov 2010;16(11):1145-1152.
- 7. Cohen RA, Moser DJ, Clark MM, et al. Neurocognitive functioning and improvement in quality of life following participation in cardiac rehabilitation. *Am J Cardiol.* May 1 1999;83(9):1374-1378.

- 8. Osowiecki DM, Cohen RA, Morrow KM, et al. Neurocognitive and psychological contributions to quality of life in HIV-1-infected women. *AIDS*. Jul 7 2000;14(10):1327-1332.
- 9. Al-Khindi T, Macdonald RL, Schweizer TA. Cognitive and functional outcome after aneurysmal subarachnoid hemorrhage. *Stroke; a journal of cerebral circulation*. Aug;41(8):e519-536.
- 10. Wadley VG, Crowe M, Marsiske M, et al. Changes in everyday function in individuals with psychometrically defined mild cognitive impairment in the Advanced Cognitive Training for Independent and Vital Elderly Study. *J Am Geriatr Soc.* Aug 2007;55(8):1192-1198.
- 11. Soderqvist A, Miedel R, Ponzer S, Tidermark J. The influence of cognitive function on outcome after a hip fracture. *The Journal of bone and joint surgery*. Oct 2006;88(10):2115-2123.
- 12. Ettenhofer ML, Hinkin CH, Castellon SA, et al. Aging, neurocognition, and medication adherence in HIV infection. *Am J Geriatr Psychiatry*. Apr 2009;17(4):281-290.
- 13. Ochner CN, Green D, van Steenburgh JJ, Kounios J, Lowe MR. Asymmetric prefrontal cortex activation in relation to markers of overeating in obese humans. *Appetite*. Aug 2009;53(1):44-49.
- 14. Reijnders J, van Heugten C, van Boxtel M. Cognitive interventions in healthy older adults and people with mild cognitive impairment: a systematic review. *Ageing Res Rev.* Jan 2013;12(1):263-275.
- 15. Li H, Li J, Li N, Li B, Wang P, Zhou T. Cognitive intervention for persons with mild cognitive impairment: A meta-analysis. *Ageing Res Rev.* Apr 2011;10(2):285-296.
- 16. Papp KV, Walsh SJ, Snyder PJ. Immediate and delayed effects of cognitive interventions in healthy elderly: a review of current literature and future directions. *Alzheimers Dement*. Jan 2009;5(1):50-60.
- 17. Ball K, Edwards JD, Ross LA. The impact of speed of processing training on cognitive and everyday functions. *The journals of gerontology. Series B, Psychological sciences and social sciences.* Jun 2007;62 Spec No 1:19-31.
- 18. Cicerone KD, Dahlberg C, Kalmar K, et al. Evidence-based cognitive rehabilitation: recommendations for clinical practice. *Arch Phys Med Rehabil.* Dec 2000;81(12):1596-1615.
- 19. Ball KK, Beard BL, Roenker DL, Miller RL, Griggs DS. Age and visual search: expanding the useful field of view. *Journal of the Optical Society of America. A, Optics and image science*. Dec 1988;5(12):2210-2219.
- 20. Ball K, Owsley C. The useful field of view test: a new technique for evaluating agerelated declines in visual function. *Journal of the American Optometric Association*. Jan 1993;64(1):71-79.
- 21. Jobe JB, Smith DM, Ball K, et al. ACTIVE: a cognitive intervention trial to promote independence in older adults. *Control Clin Trials*. Aug 2001;22(4):453-479.
- 22. Ball K, Berch DB, Helmers KF, et al. Effects of cognitive training interventions with older adults: a randomized controlled trial. *JAMA*. Nov 13 2002;288(18):2271-2281.
- 23. Edwards JD, Wadley VG, Vance DE, Wood K, Roenker DL, Ball KK. The impact of speed of processing training on cognitive and everyday performance. *Aging & mental health*. May 2005;9(3):262-271.
- 24. Willis SL, Tennstedt SL, Marsiske M, et al. Long-term effects of cognitive training on everyday functional outcomes in older adults. *JAMA*. Dec 20 2006;296(23):2805-2814.
- 25. Edwards JD, Ross LA, Ackerman ML, et al. Longitudinal predictors of driving cessation among older adults from the ACTIVE clinical trial. *The journals of gerontology. Series B, Psychological sciences and social sciences.* Jan 2008;63(1):P6-12.

- 26. Edwards JD, Myers C, Ross LA, et al. The longitudinal impact of cognitive speed of processing training on driving mobility. *The Gerontologist*. Aug 2009;49(4):485-494.
- 27. Wolinsky FD, Vander Weg MW, Martin R, et al. The effect of speed-of-processing training on depressive symptoms in ACTIVE. *The journals of gerontology. Series A, Biological sciences and medical sciences.* Apr 2009;64(4):468-472.
- 28. Ball K, Edwards JD, Ross LA, McGwin G, Jr. Cognitive training decreases motor vehicle collision involvement of older drivers. *J Am Geriatr Soc.* Nov 2010;58(11):2107-2113.
- 29. Wolinsky FD, Mahncke H, Vander Weg MW, et al. Speed of processing training protects self-rated health in older adults: enduring effects observed in the multi-site ACTIVE randomized controlled trial. *International psychogeriatrics / IPA*. May 2010;22(3):470-478.
- 30. Wolinsky FD, Vander Weg MW, Martin R, et al. Does cognitive training improve internal locus of control among older adults? *The journals of gerontology. Series B, Psychological sciences and social sciences.* Sep 2010;65(5):591-598.
- 31. Belchior P, Marsiske M, Sisco SM, et al. Video game training to improve selective visual attention in older adults. *Computers in human behavior*. Jul 1 2013;29(4):1318-1324.
- 32. Jones RN, Marsiske M, Ball K, et al. The ACTIVE cognitive training interventions and trajectories of performance among older adults. *J Aging Health*. Dec 2013;25(8 Suppl):186S-208S.
- 33. Marsiske M, Dzierzewski JM, Thomas KR, et al. Race-related disparities in 5-year cognitive level and change in untrained active participants. *J Aging Health*. Dec 2013;25(8 Suppl):103S-127S.
- 34. Ross L, Edwards, JD, Ball, K. Mobility Outcomes in ACTIVE. Paper presented at: Gerontological Society of America Meetings 2013; New Orleans, LA.
- 35. Ross LA, Edwards, J. D., & Ball, K. . Mobility Outcomes in ACTIVE. Gerontological Society of America Meetings; 2013; New Orleans, LA.
- 36. Rebok GW, Ball K, Guey LT, et al. Ten-Year Effects of the Advanced Cognitive Training for Independent and Vital Elderly Cognitive Training Trial on Cognition and Everyday Functioning in Older Adults. *J Am Geriatr Soc.* Jan 13 2014.
- 37. Edwards JD, Ruva CL, O'Brien JL, Haley CB, Lister JJ. An examination of mediators of the transfer of cognitive speed of processing training to everyday functional performance. *Psychology and aging*. Jun 2013;28(2):314-321.
- 38. Edwards JD, Hauser RA, O'Connor ML, Valdes EG, Zesiewicz TA, Uc EY. Randomized trial of cognitive speed of processing training in Parkinson disease. *Neurology*. Oct 8 2013;81(15):1284-1290.
- 39. Edwards JD, Valdes EG, Peronto C, et al. The Efficacy of InSight Cognitive Training to Improve Useful Field of View Performance: A Brief Report. *The journals of gerontology.* Series B, Psychological sciences and social sciences. Nov 8 2013.
- 40. Wolinsky FD, Unverzagt FW, Smith DM, Jones R, Wright E, Tennstedt SL. The effects of the ACTIVE cognitive training trial on clinically relevant declines in health-related quality of life. *The journals of gerontology. Series B, Psychological sciences and social sciences.* Sep 2006;61(5):S281-287.
- 41. Wolinsky FD, Vander Weg MW, Howren MB, Jones MP, Dotson MM. A randomized controlled trial of cognitive training using a visual speed of processing intervention in middle aged and older adults. *PloS one*. 2013;8(5):e61624.
- 42. Singer T, Verhaeghen P, Ghisletta P, Lindenberger U, Baltes PB. The fate of cognition in very old age: six-year longitudinal findings in the Berlin Aging Study (BASE). *Psychology and aging*. Jun 2003;18(2):318-331.
- 43. Berry AS, Zanto TP, Clapp WC, et al. The influence of perceptual training on working memory in older adults. *PloS one*. 2010;5(7):e11537.

- 44. Jaeggi SM, Buschkuehl M, Jonides J, Perrig WJ. Improving fluid intelligence with training on working memory. *Proceedings of the National Academy of Sciences of the United States of America*. May 13 2008;105(19):6829-6833.
- 45. Jaeggi SM, Buschkuehl M, Perrig WJ, Meier B. The concurrent validity of the N-back task as a working memory measure. *Memory*. May 2010;18(4):394-412.
- 46. Schneider-Garces NJ, Gordon BA, Brumback-Peltz CR, et al. Span, CRUNCH, and beyond: working memory capacity and the aging brain. *Journal of cognitive neuroscience*. Apr 2010;22(4):655-669.
- 47. Brehmer Y, Rieckmann A, Bellander M, Westerberg H, Fischer H, Backman L. Neural correlates of training-related working-memory gains in old age. *Neuroimage*. Oct 15 2011;58(4):1110-1120.
- 48. Brehmer Y, Westerberg H, Backman L. Working-memory training in younger and older adults: training gains, transfer, and maintenance. *Frontiers in human neuroscience*. 2012;6:63.
- 49. Harrison PJ. The neuropathology of schizophrenia. A critical review of the data and their interpretation. *Brain*. Apr 1999;122 ( Pt 4):593-624.
- 50. Jaeggi SM, Studer-Luethi, B., Buschkuehl, M., Su, Y. F., Jonides, J., & Perrig, W. J. . The relationship between n-back performance and matrix reasoning—Implications for training and transfer. *Intelligence*. 2010;38(6):625-635.
- 51. Jaeggi SM, Buschkuehl, M., Jonides, J., & Shah, P. Cogmed and working memory training—Current challenges and the search for underlying mechanisms. *J Appl Res Mem Cogn.* 2012;1(3):211-213.
- 52. Klingberg T. Training Working Memory. *The ADHD Report: Special Issue—Focus on Assessment.* 2006;14(1):6-8.
- 53. Coull JT, Nobre AC, Frith CD. The noradrenergic alpha2 agonist clonidine modulates behavioural and neuroanatomical correlates of human attentional orienting and alerting. *Cerebral cortex*. Jan 2001;11(1):73-84.
- 54. Heilman KM, Schwartz HD, Watson RT. Hypoarousal in patients with the neglect syndrome and emotional indifference. *Neurology*. Mar 1978;28(3):229-232.
- 55. Hjaltason H, Tegner R, Tham K, Levander M, Ericson K. Sustained attention and awareness of disability in chronic neglect. *Neuropsychologia*. Dec 1996;34(12):1229-1233.
- 56. Husain M, Shapiro K, Martin J, Kennard C. Abnormal temporal dynamics of visual attention in spatial neglect patients. *Nature*. Jan 9 1997;385(6612):154-156.
- 57. Malhotra P, Coulthard EJ, Husain M. Role of right posterior parietal cortex in maintaining attention to spatial locations over time. *Brain.* Mar 2009;132(Pt 3):645-660.
- 58. Posner MI. Measuring alertness. *Annals of the New York Academy of Sciences*. 2008:1129:193-199.
- 59. Robertson IH, Mattingley JB, Rorden C, Driver J. Phasic alerting of neglect patients overcomes their spatial deficit in visual awareness. *Nature*. Sep 10 1998;395(6698):169-172.
- 60. Sturm W, Willmes K. On the functional neuroanatomy of intrinsic and phasic alertness. *Neuroimage*. Jul 2001;14(1 Pt 2):S76-84.
- 61. Thiel CM, Zilles K, Fink GR. Cerebral correlates of alerting, orienting and reorienting of visuospatial attention: an event-related fMRI study. *Neuroimage*. Jan 2004;21(1):318-328.
- 62. Thimm M, Fink GR, Kust J, Karbe H, Sturm W. Impact of alertness training on spatial neglect: a behavioural and fMRI study. *Neuropsychologia*. 2006;44(7):1230-1246.
- 63. Woods AJ, Mennemeier M, Garcia-Rill E, et al. Improvement in arousal, visual neglect, and perception of stimulus intensity following cold pressor stimulation. *Neurocase*. 2012;18(2):115-122.

- 64. Woods AJ, Philbeck JW, Chelette K, Skinner RD, Garcia-Rill E, Mennemeier M. Cold pressor stimulation diminishes P50 amplitude in normal subjects. *Acta neurobiologiae experimentalis*. 2011;71(3):348-358.
- 65. Woods AJ, Philbeck JW, Wirtz P. Hyper-arousal decreases human visual thresholds. *PloS one.* 2013;8(4):e61415.
- 66. Degutis JM, Van Vleet TM. Tonic and phasic alertness training: a novel behavioral therapy to improve spatial and non-spatial attention in patients with hemispatial neglect. *Frontiers in human neuroscience*. 2010:4.
- 67. Van Vleet TM, Hoang-duc AK, DeGutis J, Robertson LC. Modulation of non-spatial attention and the global/local processing bias. *Neuropsychologia*. Feb 2011;49(3):352-359.
- 68. Wolinsky FD, Unverzagt FW, Smith DM, Jones R, Stoddard A, Tennstedt SL. The ACTIVE cognitive training trial and health-related quality of life: protection that lasts for 5 years. *The journals of gerontology. Series A, Biological sciences and medical sciences.* Dec 2006;61(12):1324-1329.
- 69. Antal A, Fischer T, Saiote C, et al. Transcranial electrical stimulation modifies the neuronal response to psychosocial stress exposure. *Human brain mapping*. Dec 31 2013.
- 70. Arlotti M, Rahman A, Minhas P, Bikson M. Axon terminal polarization induced by weak uniform DC electric fields: a modeling study. *Conference proceedings: ... Annual International Conference of the IEEE Engineering in Medicine and Biology Society. IEEE Engineering in Medicine and Biology Society. Conference.* 2012;2012:4575-4578.
- 71. Chrysikou EG, Hamilton RH. Noninvasive brain stimulation in the treatment of aphasia: exploring interhemispheric relationships and their implications for neurorehabilitation. *Restorative neurology and neuroscience.* 2011;29(6):375-394.
- 72. Clark VP, Coffman BA, Mayer AR, et al. TDCS guided using fMRI significantly accelerates learning to identify concealed objects. *Neuroimage*. Jan 2 2012;59(1):117-128
- 73. da Silva MC, Conti CL, Klauss J, et al. Behavioral effects of transcranial Direct Current Stimulation (tDCS) induced dorsolateral prefrontal cortex plasticity in alcohol dependence. *Journal of physiology, Paris.* Dec 2013;107(6):493-502.
- 74. Moreno-Duarte I, Morse LR, Alam M, Bikson M, Zafonte R, Fregni F. Targeted therapies using electrical and magnetic neural stimulation for the treatment of chronic pain in spinal cord injury. *Neuroimage*. Jan 15 2014;85 Pt 3:1003-1013.
- 75. Nawani H, Kalmady SV, Bose A, et al. Neural Basis of tDCS Effects on Auditory Verbal Hallucinations in Schizophrenia: A Case Report Evidence for Cortical Neuroplasticity Modulation. *The journal of ECT*. Mar 2014;30(1):e2-4.
- 76. Nitsche MA, Niehaus L, Hoffmann KT, et al. MRI study of human brain exposed to weak direct current stimulation of the frontal cortex. *Clinical neurophysiology : official journal of the International Federation of Clinical Neurophysiology.* Oct 2004;115(10):2419-2423.
- 77. Nord CL, Lally N, Charpentier CJ. Harnessing electric potential: DLPFC tDCS induces widespread brain perfusion changes. *Frontiers in systems neuroscience*. 2013;7:99.
- 78. Okano AH, Fontes EB, Montenegro RA, et al. Brain stimulation modulates the autonomic nervous system, rating of perceived exertion and performance during maximal exercise. *British journal of sports medicine.* Feb 27 2013.
- 79. Radman T, Datta A, Ramos RL, Brumberg JC, Bikson M. One-dimensional representation of a neuron in a uniform electric field. *Conference proceedings : ... Annual International Conference of the IEEE Engineering in Medicine and Biology Society. IEEE Engineering in Medicine and Biology Society. Conference.* 2009;2009:6481-6484.
- 80. Rahman A, Reato D, Arlotti M, et al. Cellular effects of acute direct current stimulation: somatic and synaptic terminal effects. *The Journal of physiology.* May 15 2013;591(Pt 10):2563-2578.
- 81. Reato D, Rahman A, Bikson M, Parra LC. Effects of weak transcranial alternating current stimulation on brain activity-a review of known mechanisms from animal studies. *Frontiers in human neuroscience*. 2013;7:687.
- 82. Sehm B, Schafer A, Kipping J, et al. Dynamic modulation of intrinsic functional connectivity by transcranial direct current stimulation. *Journal of neurophysiology*. Dec 2012;108(12):3253-3263.
- 83. Shah PP, Szaflarski JP, Allendorfer J, Hamilton RH. Induction of neuroplasticity and recovery in post-stroke aphasia by non-invasive brain stimulation. *Frontiers in human neuroscience*. 2013;7:888.
- 84. Stagg CJ, Bachtiar V, Johansen-Berg H. The role of GABA in human motor learning. *Current biology : CB.* Mar 22 2011;21(6):480-484.
- 85. Stagg CJ, Lin RL, Mezue M, et al. Widespread modulation of cerebral perfusion induced during and after transcranial direct current stimulation applied to the left dorsolateral prefrontal cortex. *J Neurosci.* Jul 10 2013;33(28):11425-11431.
- 86. Stagg CJ, Nitsche MA. Physiological basis of transcranial direct current stimulation. *The Neuroscientist: a review journal bringing neurobiology, neurology and psychiatry.* Feb 2011;17(1):37-53.
- 87. Turkeltaub PE, Benson J, Hamilton RH, Datta A, Bikson M, Coslett HB. Left lateralizing transcranial direct current stimulation improves reading efficiency. *Brain stimulation*. Jul 2012;5(3):201-207.
- 88. Woods AJ, Hamilton RH, Kranjec A, et al. Space, Time, and Causality in the Human Brain. *Neuroimage*. Feb 18 2014.
- 89. Zheng X, Alsop DC, Schlaug G. Effects of transcranial direct current stimulation (tDCS) on human regional cerebral blood flow. *Neuroimage*. Sep 1 2011;58(1):26-33.
- 90. Fregni F, Boggio PS, Santos MC, et al. Noninvasive cortical stimulation with transcranial direct current stimulation in Parkinson's disease. *Movement disorders : official journal of the Movement Disorder Society.* Oct 2006;21(10):1693-1702.
- 91. Kessler SK, Minhas P, Woods AJ, Rosen A, Gorman C, Bikson M. Dosage considerations for transcranial direct current stimulation in children: a computational modeling study. *PloS one*. 2013;8(9):e76112.
- 92. Lang N, Nitsche MA, Paulus W, Rothwell JC, Lemon RN. Effects of transcranial direct current stimulation over the human motor cortex on corticospinal and transcallosal excitability. *Experimental brain research*. Jun 2004;156(4):439-443.
- 93. Lang N, Siebner HR, Ward NS, et al. How does transcranial DC stimulation of the primary motor cortex alter regional neuronal activity in the human brain? *The European journal of neuroscience*. Jul 2005;22(2):495-504.
- 94. Liebetanz D, Nitsche MA, Tergau F, Paulus W. Pharmacological approach to the mechanisms of transcranial DC-stimulation-induced after-effects of human motor cortex excitability. *Brain.* Oct 2002;125(Pt 10):2238-2247.
- 95. Minhas P, Bikson M, Woods AJ, Rosen AR, Kessler SK. Transcranial direct current stimulation in pediatric brain: a computational modeling study. *Conference proceedings : ... Annual International Conference of the IEEE Engineering in Medicine and Biology Society. IEEE Engineering in Medicine and Biology Society. Conference.* 2012;2012:859-862.
- 96. Feng WW, Bowden MG, Kautz S. Review of transcranial direct current stimulation in poststroke recovery. *Topics in stroke rehabilitation*. Jan-Feb 2013;20(1):68-77.

- 97. Polanowska K, Seniow J. [Influence of transcranial direct current stimulation on cognitive functioning of patients with brain injury]. *Neurologia i neurochirurgia polska*. Nov-Dec 2010;44(6):580-590.
- 98. Schlaug G, Renga V. Transcranial direct current stimulation: a noninvasive tool to facilitate stroke recovery. *Expert review of medical devices*. Nov 2008;5(6):759-768.
- 99. Schlaug G, Renga V, Nair D. Transcranial direct current stimulation in stroke recovery. *Archives of neurology.* Dec 2008;65(12):1571-1576.
- 100. Berryhill ME, Jones KT. tDCS selectively improves working memory in older adults with more education. *Neuroscience letters*. Jul 19 2012;521(2):148-151.
- 101. Cerruti C, Schlaug G. Anodal transcranial direct current stimulation of the prefrontal cortex enhances complex verbal associative thought. *Journal of cognitive neuroscience*. Oct 2009;21(10):1980-1987.
- 102. Dell'Osso B, Zanoni S, Ferrucci R, et al. Transcranial direct current stimulation for the outpatient treatment of poor-responder depressed patients. *European psychiatry : the journal of the Association of European Psychiatrists*. Oct 2012;27(7):513-517.
- 103. Javadi AH, Walsh V. Transcranial direct current stimulation (tDCS) of the left dorsolateral prefrontal cortex modulates declarative memory. *Brain stimulation*. Jul 2012;5(3):231-241.
- 104. Brunoni AR, Nitsche MA, Bolognini N, et al. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. *Brain stimulation*. Jul 2012;5(3):175-195.
- 105. Cohen Kadosh R, Soskic S, Iuculano T, Kanai R, Walsh V. Modulating neuronal activity produces specific and long-lasting changes in numerical competence. *Current biology : CB.* Nov 23 2010;20(22):2016-2020.
- 106. Dockery CA, Hueckel-Weng R, Birbaumer N, Plewnia C. Enhancement of planning ability by transcranial direct current stimulation. *J Neurosci.* Jun 3 2009;29(22):7271-7277.
- 107. Hamilton RH, Chrysikou EG, Coslett B. Mechanisms of aphasia recovery after stroke and the role of noninvasive brain stimulation. *Brain and language*. Jul 2011;118(1-2):40-50.
- 108. Park SH, Seo JH, Kim YH, Ko MH. Long-term effects of transcranial direct current stimulation combined with computer-assisted cognitive training in healthy older adults. *Neuroreport*. Jan 22 2014;25(2):122-126.
- 109. Ditye T, Jacobson L, Walsh V, Lavidor M. Modulating behavioral inhibition by tDCS combined with cognitive training. *Experimental brain research*. Jun 2012;219(3):363-368
- 110. Lesniak M, Polanowska K, Seniow J, Czlonkowska A. Effects of Repeated Anodal tDCS Coupled With Cognitive Training for Patients With Severe Traumatic Brain Injury: A Pilot Randomized Controlled Trial. *The Journal of head trauma rehabilitation.* Jun 10 2013.
- 111. Li SC, Schmiedek F, Huxhold O, Rocke C, Smith J, Lindenberger U. Working memory plasticity in old age: practice gain, transfer, and maintenance. *Psychology and aging*. Dec 2008;23(4):731-742.
- 112. Martin DM, Liu R, Alonzo A, et al. Can transcranial direct current stimulation enhance outcomes from cognitive training? A randomized controlled trial in healthy participants. The international journal of neuropsychopharmacology / official scientific journal of the Collegium Internationale Neuropsychopharmacologicum. Oct 2013;16(9):1927-1936.
- 113. Kim GW, Ko MH. Facilitation of corticospinal tract excitability by transcranial direct current stimulation combined with voluntary grip exercise. *Neuroscience letters*. Aug 26 2013;548:181-184.

- 114. Krause B, Marquez-Ruiz J, Kadosh RC. The effect of transcranial direct current stimulation: a role for cortical excitation/inhibition balance? *Frontiers in human neuroscience*. 2013;7:602.
- 115. Nitsche MA, Liebetanz D, Schlitterlau A, et al. GABAergic modulation of DC stimulation-induced motor cortex excitability shifts in humans. *The European journal of neuroscience*. May 2004;19(10):2720-2726.
- 116. Ranieri F, Podda MV, Riccardi E, et al. Modulation of LTP at rat hippocampal CA3-CA1 synapses by direct current stimulation. *Journal of neurophysiology*. Apr 2012;107(7):1868-1880.
- 117. Tremblay S, Beaule V, Lepage JF, Theoret H. Anodal transcranial direct current stimulation modulates GABAB-related intracortical inhibition in the M1 of healthy individuals. *Neuroreport*. Jan 9 2013;24(1):46-50.
- 118. Stopa EG, Butala P, Salloway S, et al. Cerebral cortical arteriolar angiopathy, vascular beta-amyloid, smooth muscle actin, Braak stage, and APOE genotype. *Stroke; a journal of cerebral circulation*. Mar 2008;39(3):814-821.
- 119. Rapp MA, Schnaider-Beeri M, Purohit DP, Perl DP, Haroutunian V, Sano M. Increased neurofibrillary tangles in patients with Alzheimer disease with comorbid depression. *Am J Geriatr Psychiatry*. Feb 2008;16(2):168-174.
- 120. Mortimer JA, Gosche KM, Riley KP, Markesbery WR, Snowdon DA. Delayed recall, hippocampal volume and Alzheimer neuropathology: findings from the Nun Study. *Neurology*. Feb 10 2004;62(3):428-432.
- 121. Braak E, Griffing K, Arai K, Bohl J, Bratzke H, Braak H. Neuropathology of Alzheimer's disease: what is new since A. Alzheimer? *Eur Arch Psychiatry Clin Neurosci.* 1999;249 Suppl 3:14-22.
- 122. Thal DR, Arendt T, Waldmann G, et al. Progression of neurofibrillary changes and PHF-tau in end-stage Alzheimer's disease is different from plaque and cortical microglial pathology. *Neurobiol Aging*. Nov-Dec 1998;19(6):517-525.
- 123. Thal DR, Hartig W, Schober R. Stage-correlated distribution of type 1 and 2 dystrophic neurites in cortical and hippocampal plaques in Alzheimer's disease. *J Hirnforsch*. 1998;39(2):175-181.
- 124. Mizukami K, Grayson DR, Ikonomovic MD, Sheffield R, Armstrong DM. GABAA receptor beta 2 and beta 3 subunits mRNA in the hippocampal formation of aged human brain with Alzheimer-related neuropathology. *Brain Res Mol Brain Res.* May 1998;56(1-2):268-272.
- 125. Jellinger KA, Bancher C. Senile dementia with tangles (tangle predominant form of senile dementia). *Brain Pathol.* Apr 1998;8(2):367-376.
- 126. Nagy Z, Vatter-Bittner B, Braak H, et al. Staging of Alzheimer-type pathology: an interrater-intrarater study. *Dement Geriatr Cogn Disord*. Jul-Aug 1997;8(4):248-251.
- 127. Braak H, Braak E. Evolution of the neuropathology of Alzheimer's disease. *Acta Neurol Scand Suppl.* 1996;165:3-12.
- 128. Knopman DS, Parisi JE, Salviati A, et al. Neuropathology of cognitively normal elderly. *J Neuropathol Exp Neurol.* Nov 2003;62(11):1087-1095.
- 129. Raz N, Schmiedek F, Rodrigue KM, Kennedy KM, Lindenberger U, Lovden M. Differential brain shrinkage over 6 months shows limited association with cognitive practice. *Brain Cogn.* Jul 2013;82(2):171-180.
- 130. Fjell AM, Westlye LT, Grydeland H, et al. Critical ages in the life course of the adult brain: nonlinear subcortical aging. *Neurobiol Aging*. Oct 2013;34(10):2239-2247.
- 131. Raz N, Yang YQ, Rodrigue KM, Kennedy KM, Lindenberger U, Ghisletta P. White matter deterioration in 15 months: latent growth curve models in healthy adults. *Neurobiol Aging*. Feb 2012;33(2):429 e421-425.

- 132. Rodrigue KM, Haacke EM, Raz N. Differential effects of age and history of hypertension on regional brain volumes and iron. *Neuroimage*. Jan 15 2011;54(2):750-759.
- 133. Raz N, Ghisletta P, Rodrigue KM, Kennedy KM, Lindenberger U. Trajectories of brain aging in middle-aged and older adults: regional and individual differences. *Neuroimage*. Jun 2010;51(2):501-511.
- 134. Burgmans S, van Boxtel MP, Gronenschild EH, et al. Multiple indicators of age-related differences in cerebral white matter and the modifying effects of hypertension. *Neuroimage*. Feb 1 2010;49(3):2083-2093.
- 135. Kennedy KM, Rodrigue KM, Head D, Gunning-Dixon F, Raz N. Neuroanatomical and cognitive mediators of age-related differences in perceptual priming and learning. *Neuropsychology*. Jul 2009;23(4):475-491.
- 136. Head D, Rodrigue KM, Kennedy KM, Raz N. Neuroanatomical and cognitive mediators of age-related differences in episodic memory. *Neuropsychology*. Jul 2008;22(4):491-507.
- 137. Kennedy KM, Erickson KI, Rodrigue KM, et al. Age-related differences in regional brain volumes: a comparison of optimized voxel-based morphometry to manual volumetry. *Neurobiol Aging*. Oct 2009;30(10):1657-1676.
- 138. Raz N, Rodrigue KM, Haacke EM. Brain aging and its modifiers: insights from in vivo neuromorphometry and susceptibility weighted imaging. *Annals of the New York Academy of Sciences*. Feb 2007;1097:84-93.
- 139. Erickson KI, Colcombe SJ, Raz N, et al. Selective sparing of brain tissue in postmenopausal women receiving hormone replacement therapy. *Neurobiol Aging*. Aug-Sep 2005;26(8):1205-1213.
- 140. Raz N, Lindenberger U, Rodrigue KM, et al. Regional brain changes in aging healthy adults: general trends, individual differences and modifiers. *Cerebral cortex*. Nov 2005;15(11):1676-1689.
- 141. Raz N, Gunning-Dixon FM, Head D, Dupuis JH, Acker JD. Neuroanatomical correlates of cognitive aging: evidence from structural magnetic resonance imaging. *Neuropsychology*. Jan 1998;12(1):95-114.
- 142. Raz N, Gunning FM, Head D, et al. Selective aging of the human cerebral cortex observed in vivo: differential vulnerability of the prefrontal gray matter. *Cerebral cortex*. Apr-May 1997;7(3):268-282.
- 143. Raz N, Torres IJ, Acker JD. Age, gender, and hemispheric differences in human striatum: a quantitative review and new data from in vivo MRI morphometry. *Neurobiol Learn Mem.* Mar 1995;63(2):133-142.
- 144. Raz N, Torres IJ, Briggs SD, et al. Selective neuroanatomic abnormalities in Down's syndrome and their cognitive correlates: evidence from MRI morphometry. *Neurology*. Feb 1995;45(2):356-366.
- 145. Brickman AM, Provenzano FA, Muraskin J, et al. Regional white matter hyperintensity volume, not hippocampal atrophy, predicts incident Alzheimer disease in the community. *Archives of neurology.* Dec 2012;69(12):1621-1627.
- 146. Zimmerman ME, Brickman AM, Paul RH, et al. The relationship between frontal gray matter volume and cognition varies across the healthy adult lifespan. *Am J Geriatr Psychiatry*. Oct 2006;14(10):823-833.
- 147. Brickman AM, Habeck C, Zarahn E, Flynn J, Stern Y. Structural MRI covariance patterns associated with normal aging and neuropsychological functioning. *Neurobiol Aging*. Feb 2007;28(2):284-295.
- 148. Paul RH, Haque O, Gunstad J, et al. Subcortical hyperintensities impact cognitive function among a select subset of healthy elderly. *Arch Clin Neuropsychol.* Aug 2005;20(6):697-704.

- 149. Tate DF, Jefferson AL, Brickman AM, et al. Regional White Matter Signal Abnormalities and Cognitive Correlates Among Geriatric Patients with Treated Cardiovascular Disease. *Brain Imaging Behav.* Sep 1 2008;2(3):200-206.
- 150. Jefferson AL, Tate DF, Poppas A, et al. Lower cardiac output is associated with greater white matter hyperintensities in older adults with cardiovascular disease. *J Am Geriatr Soc.* Jul 2007;55(7):1044-1048.
- 151. Miller LA, Gunstad J, Spitznagel MB, et al. CAMTA1 T polymorphism is associated with neuropsychological test performance in older adults with cardiovascular disease. *Psychogeriatrics*. Sep 2011;11(3):135-140.
- 152. Cohen RA, Poppas A, Forman DE, et al. Vascular and cognitive functions associated with cardiovascular disease in the elderly. *J Clin Exp Neuropsychol.* Jan 2009;31(1):96-110.
- 153. Haley AP, Sweet LH, Gunstad J, et al. Verbal working memory and atherosclerosis in patients with cardiovascular disease: an fMRI study. *J Neuroimaging*. Jul 2007;17(3):227-233.
- 154. Hoth KF, Tate DF, Poppas A, et al. Endothelial function and white matter hyperintensities in older adults with cardiovascular disease. *Stroke; a journal of cerebral circulation*. Feb 2007;38(2):308-312.
- 155. Garrett KD, Browndyke JN, Whelihan W, et al. The neuropsychological profile of vascular cognitive impairment--no dementia: comparisons to patients at risk for cerebrovascular disease and vascular dementia. *Arch Clin Neuropsychol.* Sep 2004;19(6):745-757.
- 156. Alosco ML, Gunstad J, Jerskey BA, et al. The adverse effects of reduced cerebral perfusion on cognition and brain structure in older adults with cardiovascular disease. *Brain Behav.* Nov 2013;3(6):626-636.
- 157. Irani F, Sweet LH, Haley AP, et al. A fMRI Study of Verbal Working Memory, Cardiac Output, and Ejection Fraction in Elderly Patients with Cardiovascular Disease. *Brain Imaging Behav.* Dec 2009;3(4):350-357.
- 158. Haley AP, Hoth KF, Gunstad J, et al. Subjective cognitive complaints relate to white matter hyperintensities and future cognitive decline in patients with cardiovascular disease. *Am J Geriatr Psychiatry*. Nov 2009;17(11):976-985.
- 159. Gunstad J, Bausserman L, Paul RH, et al. C-reactive protein, but not homocysteine, is related to cognitive dysfunction in older adults with cardiovascular disease. *J Clin Neurosci.* Jun 2006;13(5):540-546.
- 160. Gunstad J, Cohen RA, Tate DF, et al. Blood pressure variability and white matter hyperintensities in older adults with cardiovascular disease. *Blood Press*. 2005;14(6):353-358.
- 161. Raz N, Williamson A, Gunning-Dixon F, Head D, Acker JD. Neuroanatomical and cognitive correlates of adult age differences in acquisition of a perceptual-motor skill. *Microsc Res Tech.* Oct 1 2000;51(1):85-93.
- 162. Brickman AM, Zimmerman ME, Paul RH, et al. Regional white matter and neuropsychological functioning across the adult lifespan. *Biol Psychiatry*. Sep 1 2006;60(5):444-453.
- 163. Brickman AM. Contemplating Alzheimer's disease and the contribution of white matter hyperintensities. *Curr Neurol Neurosci Rep.* Dec 2013;13(12):415.
- 164. Brickman AM, Buchsbaum MS, Shihabuddin L, Hazlett EA, Borod JC, Mohs RC. Striatal size, glucose metabolic rate, and verbal learning in normal aging. *Brain Res Cogn Brain Res*. Jun 2003;17(1):106-116.
- 165. Brickman AM, Paul RH, Cohen RA, et al. Category and letter verbal fluency across the adult lifespan: relationship to EEG theta power. *Arch Clin Neuropsychol.* Jul 2005;20(5):561-573.

- 166. Brickman AM, Schupf N, Manly JJ, et al. Brain morphology in older African Americans, Caribbean Hispanics, and whites from northern Manhattan. *Archives of neurology*. Aug 2008;65(8):1053-1061.
- 167. Brickman AM, Sneed JR, Provenzano FA, et al. Quantitative approaches for assessment of white matter hyperintensities in elderly populations. *Psychiatry Res.* Aug 30 2011;193(2):101-106.
- 168. Cohen R, Sweet LH. *Neuroimaging in Behavioral Medicine and Clinical Neuroscience*. New York, NY: Springer Publishing; 2012.
- 169. Clark US, Cohen RA, Sweet LH, et al. Effects of HIV and early life stress on amygdala morphometry and neurocognitive function. *J Int Neuropsychol Soc.* Jul 2012;18(4):657-668.
- 170. Sweet LH, Hassenstab JJ, McCaffery JM, et al. Brain response to food stimulation in obese, normal weight, and successful weight loss maintainers. *Obesity (Silver Spring)*. Nov 2012;20(11):2220-2225.
- 171. Sweet LH, Mulligan RC, Finnerty CE, et al. Effects of nicotine withdrawal on verbal working memory and associated brain response. *Psychiatry Res.* Jul 30 2010;183(1):69-74.
- 172. McCaffery JM, Haley AP, Sweet LH, et al. Differential functional magnetic resonance imaging response to food pictures in successful weight-loss maintainers relative to normal-weight and obese controls. *Am J Clin Nutr.* Oct 2009;90(4):928-934.
- 173. Browndyke JN, Paskavitz J, Sweet LH, et al. Neuroanatomical correlates of malingered memory impairment: event-related fMRI of deception on a recognition memory task. *Brain Inj.* Jun 2008;22(6):481-489.
- 174. David SP, Munafo MR, Johansen-Berg H, et al. Effects of Acute Nicotine Abstinence on Cue-elicited Ventral Striatum/Nucleus Accumbens Activation in Female Cigarette Smokers: A Functional Magnetic Resonance Imaging Study. *Brain Imaging Behav.* Dec 2007;1(3-4):43-57.
- 175. Sweet LH, Paskavitz JF, Haley AP, et al. Imaging phonological similarity effects on verbal working memory. *Neuropsychologia*. Mar 7 2008;46(4):1114-1123.
- 176. Sweet LH, Paskavitz JF, O'Connor MJ, Browndyke JN, Wellen JW, Cohen RA. FMRI correlates of the WAIS-III symbol search subtest. *J Int Neuropsychol Soc.* Jul 2005;11(4):471-476.
- 177. Sweet LH, Rao SM, Primeau M, Durgerian S, Cohen RA. Functional magnetic resonance imaging response to increased verbal working memory demands among patients with multiple sclerosis. *Human brain mapping*. Jan 2006;27(1):28-36.
- 178. Sweet LH, Rao SM, Primeau M, Mayer AR, Cohen RA. Functional magnetic resonance imaging of working memory among multiple sclerosis patients. *J Neuroimaging*. Apr 2004;14(2):150-157.
- 179. Sweet LH, Paul RH, Cohen RA, et al. Neuroimaging correlates of dementia rating scale performance at baseline and 12-month follow-up among patients with vascular dementia. *J Geriatr Psychiatry Neurol*. Dec 2003;16(4):240-244.
- 180. Davis SW, Kragel JE, Madden DJ, Cabeza R. The architecture of cross-hemispheric communication in the aging brain: linking behavior to functional and structural connectivity. *Cerebral cortex*. Jan 2012;22(1):232-242.
- 181. Madden DJ, Costello MC, Dennis NA, et al. Adult age differences in functional connectivity during executive control. *Neuroimage*. Aug 15 2010;52(2):643-657.
- 182. Davis SW, Dennis NA, Buchler NG, White LE, Madden DJ, Cabeza R. Assessing the effects of age on long white matter tracts using diffusion tensor tractography. *Neuroimage*. Jun 2009;46(2):530-541.
- 183. Davis SW, Dennis NA, Daselaar SM, Fleck MS, Cabeza R. Que PASA? The posterior-anterior shift in aging. *Cerebral cortex*. May 2008;18(5):1201-1209.

- 184. Chang L, Holt JL, Yakupov R, Jiang CS, Ernst T. Lower cognitive reserve in the aging human immunodeficiency virus-infected brain. *Neurobiol Aging*. Apr 2013;34(4):1240-1253.
- 185. Chang L, Lee P, Yiannoutsos C, et al. A multicenter In Vivo Proton MRS study of HIV-associated brain injury and the effects of aging. HIV MRS Consortium; Submitted.
- 186. Chang L, Speck O, Miller EN, et al. Neural correlates of attention and working memory deficits in HIV patients. *Neurology*. Sep 25 2001;57(6):1001-1007.
- 187. Chang L, Wong V, Nakama H, et al. Greater than age-related changes in brain diffusion of HIV patients after 1 year. *J Neuroimmune Pharmacol.* Dec 2008;3(4):265-274.
- 188. Ernst T, Chang L, Jovicich J, Ames N, Arnold S. Abnormal brain activation on functional MRI in cognitively asymptomatic HIV patients. *Neurology*. Nov 12 2002;59(9):1343-1349.
- 189. Ernst T, Itti E, Itti L, Chang L. Changes in cerebral metabolism are detected prior to perfusion changes in early HIV-CMC: A coregistered (1)H MRS and SPECT study. *J Magn Reson Imaging*. Dec 2000;12(6):859-865.
- 190. Ernst T, Yakupov R, Nakama H, et al. Declined neural efficiency in cognitively stable human immunodeficiency virus patients. *Ann Neurol.* Mar 2009;65(3):316-325.
- 191. Watanabe T, Shiino A, Akiguchi I. Absolute quantification in proton magnetic resonance spectroscopy is useful to differentiate amnesic mild cognitive impairment from Alzheimer's disease and healthy aging. *Dement Geriatr Cogn Disord*. 2010;30(1):71-77.
- 192. Ding B, Chen KM, Ling HW, et al. Diffusion tensor imaging correlates with proton magnetic resonance spectroscopy in posterior cingulate region of patients with Alzheimer's disease. *Dement Geriatr Cogn Disord*. 2008;25(3):218-225.
- 193. Metastasio A, Rinaldi P, Tarducci R, et al. Conversion of MCI to dementia: Role of proton magnetic resonance spectroscopy. *Neurobiol Aging*. Jul 2006;27(7):926-932.
- 194. Ackl N, Ising M, Schreiber YA, Atiya M, Sonntag A, Auer DP. Hippocampal metabolic abnormalities in mild cognitive impairment and Alzheimer's disease. *Neuroscience letters*. Aug 12-19 2005;384(1-2):23-28.
- 195. Modrego PJ, Fayed N, Pina MA. Conversion from mild cognitive impairment to probable Alzheimer's disease predicted by brain magnetic resonance spectroscopy. *Am J Psychiatry*. Apr 2005;162(4):667-675.
- 196. Frederick BD, Lyoo IK, Satlin A, et al. In vivo proton magnetic resonance spectroscopy of the temporal lobe in Alzheimer's disease. *Prog Neuropsychopharmacol Biol Psychiatry*. Dec 2004;28(8):1313-1322.
- 197. Pilatus U, Lais C, Rochmont Adu M, et al. Conversion to dementia in mild cognitive impairment is associated with decline of N-actylaspartate and creatine as revealed by magnetic resonance spectroscopy. *Psychiatry Res.* Jul 15 2009;173(1):1-7.
- 198. Waldman AD, Rai GS. The relationship between cognitive impairment and in vivo metabolite ratios in patients with clinical Alzheimer's disease and vascular dementia: a proton magnetic resonance spectroscopy study. *Neuroradiology*. Aug 2003;45(8):507-512.
- 199. Pagonabarraga J, Gomez-Anson B, Rotger R, et al. Spectroscopic changes associated with mild cognitive impairment and dementia in Parkinson's disease. *Dement Geriatr Cogn Disord*. 2012;34(5-6):312-318.
- 200. Gasparovic C, Prestopnik J, Thompson J, et al. 1H-MR spectroscopy metabolite levels correlate with executive function in vascular cognitive impairment. *J Neurol Neurosurg Psychiatry*. Jul 2013;84(7):715-721.
- 201. Wang S, Yuan J, Guo X, et al. Neurochemical correlates of cognitive dysfunction in patients with leukoaraiosis: a proton magnetic resonance spectroscopy study. *Neurol Res.* Dec 2012;34(10):989-997.

- 202. Griffith HR, Stewart CC, den Hollander JA. Proton magnetic resonance spectroscopy in dementias and mild cognitive impairment. *Int Rev Neurobiol.* 2009;84:105-131.
- 203. Ross AJ, Sachdev PS, Wen W, Valenzuela MJ, Brodaty H. 1H MRS in stroke patients with and without cognitive impairment. *Neurobiol Aging*. Jun 2005;26(6):873-882.
- 204. Chang L, Lee PL, Yiannoutsos CT, et al. A multicenter in vivo proton-MRS study of HIV-associated dementia and its relationship to age. *Neuroimage*. Dec 2004;23(4):1336-1347.
- 205. Lee PL, Yiannoutsos CT, Ernst T, et al. A multi-center 1H MRS study of the AIDS dementia complex: validation and preliminary analysis. *J Magn Reson Imaging*. Jun 2003;17(6):625-633.
- 206. Yiannoutsos CT, Ernst T, Chang L, et al. Regional patterns of brain metabolites in AIDS dementia complex. *Neuroimage*. Nov 2004;23(3):928-935.
- 207. Hua X, Boyle CP, Harezlak J, et al. Disrupted cerebral metabolite levels and lower nadir CD4 + counts are linked to brain volume deficits in 210 HIV-infected patients on stable treatment. *Neuroimage Clin.* 2013;3:132-142.
- 208. Harezlak J, Buchthal S, Taylor M, et al. Persistence of HIV-associated cognitive impairment, inflammation, and neuronal injury in era of highly active antiretroviral treatment. *AIDS*. Mar 13 2011;25(5):625-633.
- 209. Cohen RA, Harezlak J, Gongvatana A, et al. Cerebral metabolite abnormalities in human immunodeficiency virus are associated with cortical and subcortical volumes. *Journal of neurovirology*. Nov 2010;16(6):435-444.
- 210. Paul RH, Ernst T, Brickman AM, et al. Relative sensitivity of magnetic resonance spectroscopy and quantitative magnetic resonance imaging to cognitive function among nondemented individuals infected with HIV. *J Int Neuropsychol Soc.* Sep 2008;14(5):725-733.
- 211. Paul RH, Gunstad J, Cooper N, et al. Cross-cultural assessment of neuropsychological performance and electrical brain function measures: additional validation of an international brain database. *Int J Neurosci.* Apr 2007;117(4):549-568.
- 212. Watanabe M, Maemura K, Kanbara K, Tamayama T, Hayasaki H. GABA and GABA receptors in the central nervous system and other organs. *Int Rev Cytol.* 2002;213:1-47.
- 213. Szabadics J, Varga C, Molnar G, Olah S, Barzo P, Tamas G. Excitatory effect of GABAergic axo-axonic cells in cortical microcircuits. *Science*. Jan 13 2006;311(5758):233-235.
- 214. Foster TC, Sharrow KM, Kumar A, Masse J. Interaction of age and chronic estradiol replacement on memory and markers of brain aging. *Neurobiol Aging*. Oct 2003;24(6):839-852.
- 215. Foster TC, Kumar A. Calcium dysregulation in the aging brain. *The Neuroscientist : a review journal bringing neurobiology, neurology and psychiatry.* Aug 2002;8(4):297-301.
- 216. Foster TC, Sharrow KM, Masse JR, Norris CM, Kumar A. Calcineurin links Ca2+ dysregulation with brain aging. *J Neurosci.* Jun 1 2001;21(11):4066-4073.
- 217. Foster TC. Involvement of hippocampal synaptic plasticity in age-related memory decline. *Brain Res Brain Res Rev.* Nov 1999;30(3):236-249.
- 218. Foster TC, Norris CM. Age-associated changes in Ca(2+)-dependent processes: relation to hippocampal synaptic plasticity. *Hippocampus*. 1997;7(6):602-612.
- 219. Baumgartner BJ, Harvey RJ, Darlison MG, Barnes EM, Jr. Developmental up-regulation and agonist-dependent down-regulation of GABAA receptor subunit mRNAs in chick cortical neurons. *Brain Res Mol Brain Res*. Oct 1994;26(1-2):9-17.
- 220. Green EJ, Barnes CA, McNaughton BL. Behavioral state dependence of homo- and hetero-synaptic modulation of dentate gyrus excitability. *Experimental brain research*. 1993;93(1):55-65.

- 221. Mizumori SJ, Barnes CA, McNaughton BL. Differential effects of age on subpopulations of hippocampal theta cells. *Neurobiol Aging*. Nov-Dec 1992;13(6):673-679.
- 222. Burke SN, Barnes CA. Senescent synapses and hippocampal circuit dynamics. *Trends Neurosci.* Mar 2010;33(3):153-161.
- 223. Burke SN, Maurer AP, Yang Z, Navratilova Z, Barnes CA. Glutamate receptor-mediated restoration of experience-dependent place field expansion plasticity in aged rats. *Behav Neurosci.* Jun 2008;122(3):535-548.
- 224. Barnes J, Hinkley L, Masters S, Boubert L. Visual memory transformations in dyslexia. *Percept Mot Skills.* Jun 2007;104(3 Pt 1):881-891.
- 225. Barnes P, Good M. Impaired Pavlovian cued fear conditioning in Tg2576 mice expressing a human mutant amyloid precursor protein gene. *Behav Brain Res.* Feb 10 2005;157(1):107-117.
- 226. Barnes DE, Tager IB, Satariano WA, Yaffe K. The relationship between literacy and cognition in well-educated elders. *The journals of gerontology. Series A, Biological sciences and medical sciences*. Apr 2004;59(4):390-395.
- 227. Barnes CA. Long-term potentiation and the ageing brain. *Philos Trans R Soc Lond B Biol Sci.* Apr 29 2003;358(1432):765-772.
- 228. Barnes CA, Rao G, Orr G. Age-related decrease in the Schaffer collateral-evoked EPSP in awake, freely behaving rats. *Neural Plast.* 2000;7(3):167-178.
- 229. Barnes CA, Rao G, Houston FP. LTP induction threshold change in old rats at the perforant path--granule cell synapse. *Neurobiol Aging*. Sep-Oct 2000;21(5):613-620.
- 230. Barnes CA, Rao G, Shen J. Age-related decrease in the N-methyl-D-aspartateR-mediated excitatory postsynaptic potential in hippocampal region CA1. *Neurobiol Aging*. Jul-Aug 1997;18(4):445-452.
- 231. Rao G, Barnes CA, McNaughton BL. Effects of age on L-glutamate-induced depolarization in three hippocampal subfields. *Neurobiol Aging*. Jan-Feb 1993;14(1):27-33.
- 232. Nelson HE, Pantelis C, Carruthers K, Speller J, Baxendale S, Barnes TR. Cognitive functioning and symptomatology in chronic schizophrenia. *Psychol Med.* May 1990;20(2):357-365.
- 233. Barnes CA. Effects of aging on the dynamics of information processing and synaptic weight changes in the mammalian hippocampus. *Prog Brain Res.* 1990;86:89-104.
- 234. Barnes CA. Aging and the physiology of spatial memory. *Neurobiol Aging*. Sep-Dec 1988;9(5-6):563-568.
- 235. Barnes CA. Memory deficits associated with senescence: a neurophysiological and behavioral study in the rat. *J Comp Physiol Psychol.* Feb 1979;93(1):74-104.
- 236. Alexander GE, Ryan L, Bowers D, et al. Characterizing cognitive aging in humans with links to animal models. *Front Aging Neurosci.* 2012;4:21.
- 237. Bizon JL, Foster TC, Alexander GE, Glisky EL. Characterizing cognitive aging of working memory and executive function in animal models. *Front Aging Neurosci.* 2012;4:19.
- 238. Roberson ED, Defazio RA, Barnes CA, et al. Challenges and opportunities for characterizing cognitive aging across species. *Front Aging Neurosci.* 2012;4:6.
- 239. Nilsen LH, Melo TM, Saether O, Witter MP, Sonnewald U. Altered neurochemical profile in the McGill-R-Thy1-APP rat model of Alzheimer's disease: a longitudinal in vivo 1 H MRS study. *J Neurochem*. Nov 2012;123(4):532-541.
- 240. Martin WR. MR spectroscopy in neurodegenerative disease. *Mol Imaging Biol.* Jul-Aug 2007;9(4):196-203.
- 241. Broccardo C, Nieoullon V, Amin R, et al. ABCA2 is a marker of neural progenitors and neuronal subsets in the adult rodent brain. *J Neurochem*. Apr 2006;97(2):345-355.

- 242. Wang H, Lian K, Han B, et al. Age-Related Alterations in the Metabolic Profile in the Hippocampus of the Senescence-Accelerated Mouse Prone 8: A Spontaneous Alzheimer's Disease Mouse Model. *J Alzheimers Dis.* Nov 27 2013.
- 243. Paul SM, Doherty JJ, Robichaud AJ, et al. The major brain cholesterol metabolite 24(S)-hydroxycholesterol is a potent allosteric modulator of N-methyl-D-aspartate receptors. *J Neurosci.* Oct 30 2013;33(44):17290-17300.
- 244. Nilsen LH, Rae C, Ittner LM, Gotz J, Sonnewald U. Glutamate metabolism is impaired in transgenic mice with tau hyperphosphorylation. *J Cereb Blood Flow Metab*. May 2013;33(5):684-691.
- 245. Ferchmin PA, Perez D, Castro Alvarez W, Penzo MA, Maldonado HM, Eterovic VA. gamma-Aminobutyric acid type A receptor inhibition triggers a nicotinic neuroprotective mechanism. *J Neurosci Res.* Mar 2013;91(3):416-425.
- 246. Koh MT, Rosenzweig-Lipson S, Gallagher M. Selective GABA(A) alpha5 positive allosteric modulators improve cognitive function in aged rats with memory impairment. *Neuropharmacology.* Jan 2013;64:145-152.
- 247. Leon-Espinosa G, DeFelipe J, Munoz A. Effects of amyloid-beta plaque proximity on the axon initial segment of pyramidal cells. *J Alzheimers Dis.* 2012;29(4):841-852.
- 248. Krantic S, Isorce N, Mechawar N, et al. Hippocampal GABAergic neurons are susceptible to amyloid-beta toxicity in vitro and are decreased in number in the Alzheimer's disease TgCRND8 mouse model. *J Alzheimers Dis.* 2012;29(2):293-308.
- 249. Poil SS, Jansen R, van Aerde K, et al. Fast network oscillations in vitro exhibit a slow decay of temporal auto-correlations. *The European journal of neuroscience*. Aug 2011;34(3):394-403.
- 250. Li G, Bien-Ly N, Andrews-Zwilling Y, et al. GABAergic interneuron dysfunction impairs hippocampal neurogenesis in adult apolipoprotein E4 knockin mice. *Cell Stem Cell*. Dec 4 2009;5(6):634-645.
- 251. Rangel A, Madronal N, Gruart A, et al. Regulation of GABA(A) and glutamate receptor expression, synaptic facilitation and long-term potentiation in the hippocampus of prion mutant mice. *PloS one*. 2009;4(10):e7592.
- 252. Molinaro G, Battaglia G, Riozzi B, et al. Memantine treatment reduces the expression of the K(+)/Cl(-) cotransporter KCC2 in the hippocampus and cerebral cortex, and attenuates behavioural responses mediated by GABA(A) receptor activation in mice. *Brain Res.* Apr 10 2009;1265:75-79.
- 253. Matsuyama S, Taniguchi T, Kadoyama K, Matsumoto A. Long-term potentiation-like facilitation through GABAA receptor blockade in the mouse dentate gyrus in vivo. *Neuroreport.* Dec 3 2008;19(18):1809-1813.
- 254. Yuk DY, Lee YK, Nam SY, et al. Reduced anxiety in the mice expressing mutant (N141I) presenilin 2. *J Neurosci Res.* Feb 2009;87(2):522-531.
- 255. Albuquerque EX, Pereira EF, Mike A, Eisenberg HM, Maelicke A, Alkondon M. Neuronal nicotinic receptors in synaptic functions in humans and rats: physiological and clinical relevance. *Behav Brain Res.* Aug 2000;113(1-2):131-141.
- 256. Alkondon M, Pereira EF, Yu P, et al. Targeted deletion of the kynurenine aminotransferase ii gene reveals a critical role of endogenous kynurenic acid in the regulation of synaptic transmission via alpha7 nicotinic receptors in the hippocampus. *J Neurosci.* May 12 2004;24(19):4635-4648.
- 257. Edgar PF, Schonberger SJ, Dean B, Faull RL, Kydd R, Cooper GJ. A comparative proteome analysis of hippocampal tissue from schizophrenic and Alzheimer's disease individuals. *Mol Psychiatry*. Mar 1999;4(2):173-178.
- 258. Griguoli M, Cherubini E. Regulation of hippocampal inhibitory circuits by nicotinic acetylcholine receptors. *The Journal of physiology.* Feb 15 2012;590(Pt 4):655-666.

- 259. Uehara T, Sumiyoshi T, Hattori H, et al. T-817MA, a novel neurotrophic agent, ameliorates loss of GABAergic parvalbumin-positive neurons and sensorimotor gating deficits in rats transiently exposed to MK-801 in the neonatal period. *J Psychiatr Res.* May 2012;46(5):622-629.
- 260. Tao R, Li C, Newburn EN, et al. Transcript-specific associations of SLC12A5 (KCC2) in human prefrontal cortex with development, schizophrenia, and affective disorders. *J Neurosci.* Apr 11 2012;32(15):5216-5222.
- 261. Pattwell SS, Bath KG, Perez-Castro R, Lee FS, Chao MV, Ninan I. The BDNF Val66Met polymorphism impairs synaptic transmission and plasticity in the infralimbic medial prefrontal cortex. *J Neurosci.* Feb 15 2012;32(7):2410-2421.
- 262. Vinkers CH, Oosting RS, van Bogaert MJ, Olivier B, Groenink L. Early-life blockade of 5-HT(1A) receptors alters adult anxiety behavior and benzodiazepine sensitivity. *Biol Psychiatry*. Feb 15 2010;67(4):309-316.
- 263. Miczek KA, Yap JJ, Covington HE, 3rd. Social stress, therapeutics and drug abuse: preclinical models of escalated and depressed intake. *Pharmacol Ther.* Nov 2008;120(2):102-128.
- 264. Hoschl C, Hajek T. Hippocampal damage mediated by corticosteroids--a neuropsychiatric research challenge. *Eur Arch Psychiatry Clin Neurosci.* 2001;251 Suppl 2:II81-88.
- 265. Motohashi N, Ikawa K, Kariya T. GABAB receptors are up-regulated by chronic treatment with lithium or carbamazepine. GABA hypothesis of affective disorders? *Eur J Pharmacol.* Jul 4 1989;166(1):95-99.
- 266. Martin P, Pichat P, Massol J, Soubrie P, Lloyd KG, Puech AJ. Decreased GABA B receptors in helpless rats: reversal by tricyclic antidepressants. *Neuropsychobiology*. 1989;22(4):220-224.
- 267. Lloyd KG, Morselli PL, Bartholini G. GABA and affective disorders. *Med Biol.* 1987;65(2-3):159-165.
- 268. Long Z, Li XR, Xu J, et al. Thalamic GABA Predicts Fine Motor Performance in Manganese-Exposed Smelter Workers. *PloS one.* 2014;9(2):e88220.
- 269. Mullins PG, McGonigle DJ, O'Gorman RL, et al. Current practice in the use of MEGA-PRESS spectroscopy for the detection of GABA. *Neuroimage*. Feb 1 2014;86:43-52.
- 270. Shaw A, Brealy J, Richardson H, et al. Marked reductions in visual evoked responses but not gamma-aminobutyric acid concentrations or gamma-band measures in remitted depression. *Biol Psychiatry*. Apr 1 2013;73(7):691-698.
- 271. Foerster BR, Callaghan BC, Petrou M, Edden RA, Chenevert TL, Feldman EL. Decreased motor cortex gamma-aminobutyric acid in amyotrophic lateral sclerosis. *Neurology.* May 15 2012;78(20):1596-1600.
- 272. Stone JM, Dietrich C, Edden R, et al. Ketamine effects on brain GABA and glutamate levels with 1H-MRS: relationship to ketamine-induced psychopathology. *Mol Psychiatry*. Jul 2012;17(7):664-665.
- 273. Dydak U, Jiang YM, Long LL, et al. In vivo measurement of brain GABA concentrations by magnetic resonance spectroscopy in smelters occupationally exposed to manganese. *Environ Health Perspect.* Feb 2011;119(2):219-224.
- 274. Edden RA, Puts NA, Barker PB. Macromolecule-suppressed GABA-edited magnetic resonance spectroscopy at 3T. *Magn Reson Med.* Sep 2012;68(3):657-661.
- 275. Edden RA, Crocetti D, Zhu H, Gilbert DL, Mostofsky SH. Reduced GABA concentration in attention-deficit/hyperactivity disorder. *Arch Gen Psychiatry*. Jul 2012;69(7):750-753.
- 276. Michels L, Martin E, Klaver P, et al. Frontal GABA levels change during working memory. *PloS one.* 2012;7(4):e31933.

- 277. Edden RA, Intrapiromkul J, Zhu H, Cheng Y, Barker PB. Measuring T2 in vivo with J-difference editing: application to GABA at 3 Tesla. *J Magn Reson Imaging*. Jan 2012;35(1):229-234.
- 278. Edden RA, Barker PB. If J doesn't evolve, it won't J-resolve: J-PRESS with bandwidth-limited refocusing pulses. *Magn Reson Med.* Jun 2011;65(6):1509-1514.
- 279. Sisco SM, Marsiske M, Gross AL, Rebok GW. The influence of cognitive training on older adults' recall for short stories. *J Aging Health*. Dec 2013;25(8 Suppl):230S-248S.
- 280. Payne BR, Gross AL, Parisi JM, et al. Modelling longitudinal changes in older adults' memory for spoken discourse: Findings from the ACTIVE cohort. *Memory*. Dec 4 2013.
- 281. Merzenich M. POSIT Science. 2014; http://www.positscience.com.
- 282. Nadeau SE, Wu SS. CIMT as a behavioral engine in research on physiological adjuvants to neurorehabilitation: the challenge of merging animal and human research. *NeuroRehabilitation*. 2006;21(2):107-130.
- 283. Batsikadze G, Moliadze V, Paulus W, Kuo MF, Nitsche MA. Partially non-linear stimulation intensity-dependent effects of direct current stimulation on motor cortex excitability in humans. *The Journal of physiology.* Apr 1 2013;591(Pt 7):1987-2000.
- 284. Trahan DE, Larrabee GJ, Quintana JW. Visual recognition memory in normal adults and patients with unilateral vascular lesions. *J Clin Exp Neuropsychol.* Dec 1990;12(6):857-872.
- 285. Larrabee GJ, Trahan DE, Curtiss G. Construct validity of the Continuous Visual Memory Test. *Arch Clin Neuropsychol*. Oct 1992;7(5):395-405.
- 286. Paolo AM, Troster AI, Ryan JJ. Test-retest stability of the Continuous Visual Memory Test in elderly persons. *Arch Clin Neuropsychol.* Oct 1998;13(7):617-621.
- 287. Paolo AM, Troster AI, Ryan JJ. Continuous Visual Memory Test performance in healthy persons 60 to 94 years of age. *Arch Clin Neuropsychol*. May 1998;13(4):333-337.
- 288. Snitz BE, Roman DD, Beniak TE. Efficacy of the Continuous Visual Memory Test in lateralizing temporal lobe dysfunction in chronic complex-partial epilepsy. *J Clin Exp Neuropsychol*. Oct 1996;18(5):747-754.
- 289. Hall S, Pinkston SL, Szalda-Petree AC, Coronis AR. The performance of healthy older adults on the Continuous Visual Memory Test and the Visual-Motor Integration Test: preliminary findings. *J Clin Psychol*. Jul 1996;52(4):449-454.
- 290. Harker KT, Connolly JF. Assessment of visual working memory using event-related potentials. *Clinical neurophysiology: official journal of the International Federation of Clinical Neurophysiology.* Nov 2007;118(11):2479-2488.
- 291. Banos JH, Dickson AL, Greer T. A computer-assisted administration of the Continuous Visual Memory Test. *Clin Neuropsychol.* Dec 2001;15(4):551-555.
- 292. Retzlaff PD, Morris GL. Event-related potentials during the Continuous Visual Memory Test. *J Clin Psychol.* Jan 1996;52(1):43-47.
- 293. Woods AJ, Hamilton, et al., . Space, time, and causaltiy in the human brain. *Neuroimage*. 2014;in press.
- 294. Woods AJ, Lehet M, Chatterjee A. Context modulates the contribution of time and space in causal inference. *Front Psychol.* 2012;3:371.
- 295. Provencher SW. Automatic quantitation of localized in vivo 1H spectra with LCModel. *NMR in biomedicine*. Jun 2001;14(4):260-264.
- 296. Fischl B, Dale AM. Measuring the thickness of the human cerebral cortex from magnetic resonance images. *Proceedings of the National Academy of Sciences of the United States of America*. Sep 26 2000;97(20):11050-11055.
- 297. Fischl B, Sereno MI, Dale AM. Cortical surface-based analysis. II: Inflation, flattening, and a surface-based coordinate system. *Neuroimage*. Feb 1999;9(2):195-207.
- 298. Fischl B, Sereno MI, Tootell RB, Dale AM. High-resolution intersubject averaging and a coordinate system for the cortical surface. *Human brain mapping*. 1999;8(4):272-284.

- 299. Andrade KC, Pontes-Neto OM, Leite JP, Santos AC, Baffa O, de Araujo DB. Quantitative aspects of brain perfusion dynamic induced by BOLD fMRI. *Arq Neuropsiguiatr.* Dec 2006;64(4):895-898.
- 300. Leoni RF, Mazzeto-Betti KC, Andrade KC, de Araujo DB. Quantitative evaluation of hemodynamic response after hypercapnia among different brain territories by fMRI. *Neuroimage*. Jul 15 2008;41(4):1192-1198.
- 301. Kim SG, Rostrup E, Larsson HB, Ogawa S, Paulson OB. Determination of relative CMRO2 from CBF and BOLD changes: significant increase of oxygen consumption rate during visual stimulation. *Magn Reson Med.* Jun 1999;41(6):1152-1161.
- 302. Kastrup A, Kruger G, Glover GH, Neumann-Haefelin T, Moseley ME. Regional variability of cerebral blood oxygenation response to hypercapnia. *Neuroimage*. Dec 1999;10(6):675-681.
- 303. Posse S, Kemna LJ, Elghahwagi B, Wiese S, Kiselev VG. Effect of graded hypo- and hypercapnia on fMRI contrast in visual cortex: quantification of T(\*)(2) changes by multiecho EPI. *Magn Reson Med.* Aug 2001;46(2):264-271.
- 304. Lezak MD. Neuropsychological assessment in behavioral toxicology--developing techniques and interpretative issues. *Scandinavian journal of work, environment & health.* 1984;10 Suppl 1:25-29.
- 305. DiGirolamo GJ, Kramer AF, Barad V, et al. General and task-specific frontal lobe recruitment in older adults during executive processes: a fMRI investigation of task-switching. *Neuroreport*. Jul 3 2001;12(9):2065-2071.
- 306. Gross AL, Rebok GW, Brandt J, Tommet D, Marsiske M, Jones RN. Modeling learning and memory using verbal learning tests: results from ACTIVE. *The journals of gerontology. Series B, Psychological sciences and social sciences.* Mar 2013;68(2):153-167.
- 307. Gunstad J, Cohen RA, Paul RH, Luyster FS, Gordon E. Age effects in time estimation: relationship to frontal brain morphometry. *Journal of integrative neuroscience*. Mar 2006;5(1):75-87.
- 308. Jones RN, Rosenberg AL, Morris JN, et al. A growth curve model of learning acquisition among cognitively normal older adults. *Experimental aging research*. Jul-Sep 2005;31(3):291-312.
- 309. Okonkwo OC, Cohen RA, Gunstad J, Tremont G, Alosco ML, Poppas A. Longitudinal trajectories of cognitive decline among older adults with cardiovascular disease. *Cerebrovasc Dis.* 2010;30(4):362-373.
- 310. Paul RH, Brickman AM, Cohen RA, et al. Cognitive status of young and older cigarette smokers: data from the international brain database. *J Clin Neurosci.* May 2006;13(4):457-465.
- 311. Roller CA, Cohen HS, Kimball KT, Bloomberg JJ. Effects of normal aging on visuo-motor plasticity. *Neurobiol Aging*. Jan-Feb 2002;23(1):117-123.
- 312. Woods AJ, Mark VW, Pitts AC, Mennemeier M. Pervasive cognitive impairment in acute rehabilitation inpatients without brain injury. *PM & R : the journal of injury, function, and rehabilitation.* May 2011;3(5):426-432; quiz 432.
- 313. Zimerman M, Nitsch M, Giraux P, Gerloff C, Cohen LG, Hummel FC. Neuroenhancement of the aging brain: restoring skill acquisition in old subjects. *Ann Neurol.* Jan 2013;73(1):10-15.
- 314. Zlatar ZZ, Towler S, McGregor KM, et al. Functional language networks in sedentary and physically active older adults. *J Int Neuropsychol Soc.* Jul 2013;19(6):625-634.
- 315. Taha J, Czaja SJ, Sharit J, Morrow DG. Factors affecting usage of a personal health record (PHR) to manage health. *Psychology and aging.* Dec 2013;28(4):1124-1139.

- 316. Sharit J, Czaja SJ, Nair S, Lee CC. Effects of age, speech rate, and environmental support in using telephone voice menu systems. *Hum Factors*. Summer 2003;45(2):234-251.
- 317. Baecke JA, Burema J, Frijters JE. A short questionnaire for the measurement of habitual physical activity in epidemiological studies. *Am J Clin Nutr.* Nov 1982;36(5):936-942.
- 318. Richardson MT, Ainsworth BE, Wu HC, Jacobs DR, Jr., Leon AS. Ability of the Atherosclerosis Risk in Communities (ARIC)/Baecke Questionnaire to assess leisure-time physical activity. *International journal of epidemiology*. Aug 1995;24(4):685-693.
- 319. Philippaerts RM, Westerterp KR, Lefevre J. Doubly labelled water validation of three physical activity questionnaires. *International journal of sports medicine*. Jul 1999;20(5):284-289.
- 320. Philippaerts RM, Lefevre J. Reliability and validity of three physical activity questionnaires in Flemish males. *American journal of epidemiology*. May 15 1998;147(10):982-990.
- 321. Cella D, Riley W, Stone A, et al. The Patient-Reported Outcomes Measurement Information System (PROMIS) developed and tested its first wave of adult self-reported health outcome item banks: 2005-2008. *Journal of clinical epidemiology.* Nov 2010;63(11):1179-1194.
- 322. Magasi S, Ryan G, Revicki D, et al. Content validity of patient-reported outcome measures: perspectives from a PROMIS meeting. *Quality of life research: an international journal of quality of life aspects of treatment, care and rehabilitation.* Jun 2012;21(5):739-746.
- 323. Tucker CA, Cieza A, Riley AW, et al. Concept Analysis of the Patient Reported Outcomes Measurement Information System (PROMIS) and the International Classification of Functioning, Disability and Health (ICF). Quality of life research: an international journal of quality of life aspects of treatment, care and rehabilitation. Feb 6 2014.
- 324. Reeve BB, Hays RD, Bjorner JB, et al. Psychometric evaluation and calibration of health-related quality of life item banks: plans for the Patient-Reported Outcomes Measurement Information System (PROMIS). *Medical care*. May 2007;45(5 Suppl 1):S22-31.